#### CONFIDENTIAL

## GlaxoSmithKline group of companies

PHI201754

#### TITLE PAGE

**Division**: Worldwide Development **Information Type**: Clinical Protocol

**Title:** A 52-week, Phase III, double-blind, active-controlled, parallel-group, multi-center study to evaluate efficacy and safety of daprodustat compared to darbepoetin alfa in Japanese hemodialysis-dependent subjects with anemia associated with chronic kidney disease who are currently ESA users.

**Compound Number:** Daprodustat

**Development Phase** III

Effective Date: 19-Jul-2017

**Protocol Amendment Number:** 02

## Author(s):

PPD

PPD

## **Revision Chronology:**

| GlaxoSmithKline Document<br>Number | Date | Version |
|------------------------------------|-------------|---------------|
| 2015N266251_00 | 19-JUL-2016 | First version |
| 2015N266251_01 | 08-MAR-2017 | Amendment 01 |

Clarification of the timing of eligibility assessment regarding exclusion criteria, addition of the prohibited medication, and correction of adverse events of special interest

| 2015N266251 02 | 19-JUL-2017 | Amendment 02 |
|-------------------|-------------|--------------|
| 1 201311200231 02 | 17-JUL-2017 | Amenument 02 |

Change for definition of screen failures, clarification of the withdrawal/dropout criteria for prohibited medication, clarification of definition of overdose of daprodustat, update of AESI, addition of details of sensitivity analyses for primary efficacy analysis and description adjustment, update of risk assessment (Appendix 2), and correction of erroneous description

Copyright 2016 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

| 20 | 151 | 126 | 625 | 1 | 02 |
|----|-----|-----|-----|---|----|

# **CONFIDENTIAL**

PHI201754

| <b>Sponsor Signatory:</b> |
|---------------------------|
|---------------------------|

Kihito Takahashi Date

Director,

Japan Development and Medical Affairs (JDMA),

GlaxoSmithKline K. K.

The IMMS document approved is as follows:

Unique ID: 090033ec8416fd56

System Version:1.0

Effective Date: 19 Jul 2017

# MEDICAL MONITOR/SPONSOR INFORMATION PAGE

# **Medical Monitor/SAE Contact Information:**

| Role | Name | Day Time<br>Phone<br>Number | Fax Number | Site Address |
|---|---|---|---|---|
| Medical Monitor | PPD<br>M.D., Ph.D. | PPD | | GlaxoSmithKline K.K.<br>6-15, Sendagaya 4-chome,<br>Shibuya-ku, Tokyo 151-8566<br>JAPAN |
| SAE contact information | Person in charge<br>of daprodustat<br>Clinical<br>Operations dept. | | | GlaxoSmithKline K.K.<br>6-15, Sendagaya 4-chome,<br>Shibuya-ku, Tokyo 151-8566<br>JAPAN |

# **Emergency Contact**

Emergency Contact (Mon to Fri 10am to 6pm, except for national holiday and year-end and New Year holidays)

Person in charge of daprodustat, Clinical Operations dept. R&D, Glaxo Smith Kline K.K

TEL: PPD FAX:

Emergency Contact at night and holiday (Mon to Fri 6pm to 10am, Sat, Sun, national holiday and year-end and New Year holidays)

BI Medical Inc.

Responsible Person: PPD
TEL: PPD (toll free)
FAX: (toll free)

# **Sponsor Legal Registered Address:**

6-15, Sendagaya 4-chome, Shibuya-ku, Tokyo 151-8566 JAPAN

# **INVESTIGATOR PROTOCOL AGREEMENT PAGE**

- I confirm agreement to conduct the study in compliance with the protocol and the amended content.
- I acknowledge that I am responsible for overall study conduct. I agree to personally conduct or supervise the described study.
- I agree to ensure that all associates, colleagues and employees assisting in the conduct of the study are informed about their obligations. Mechanisms are in place to ensure that site staff receives the appropriate information throughout the study.

•

| Investigator Name: | |
|------------------------|------|
| Investigator Signature | Date |

# **TABLE OF CONTENTS**

| | | | | Page |
|---|---|---|---|---|
| 1. | PR | отос | OL SYNOPSIS FOR STUDY PHI201754 | 9 |
| 2. | INT | TRODU | ICTION | 13 |
| | 2.1. | Stud | dy Rationale | 13 |
| | 2.2. | Bacl | kground | 13 |
| 3. | OB | BJECTI | VES AND ENDPOINTS | 14 |
| 4. | ST | UDY D | ESIGN | 16 |
| | 4.1. | Ove | rall Design | 16 |
| | 4.2. | Trea | tment Groups and Study Periods | 16 |
| | 4.3. | Stud | dy Subjects and Number of Subjects | 17 |
| | 4.4. | Ratio | onale for Study Design | 17 |
| | 4.5. | Ratio | onale for Dose Levels | 18 |
| | 4.6. | Ben | efit: Risk Assessment | 19 |
| | 4.6 | 5.1. | Risk Assessment | 19 |
| | 4.6 | 5.2. | Benefit Assessment | 19 |
| | 4.6 | 5.3. | Overall Benefit: Risk Conclusion | 20 |
| 5. | SU | IBJEC1 | SELECTION AND WITHDRAWAL CRITERIA | 21 |
| | 5.1. | Inclu | usion Criteria | 21 |
| | 5.2. | Excl | lusion Criteria | 22 |
| | 5.3. | Scre | eening Failures | 23 |
| | 5.4. | Pern | nanent discontinuation of study treatment and study withdrawal | 24 |
| | 5.4 | l.1. | Liver Chemistry Stopping Criteria | 25 |
| | 5 | 5.4.1.1. | Study Treatment Restart or Rechallenge | 26 |
| | 5.5. | Subj | ject and Study Completion | 26 |
| 6. | ST | UDY T | REATMENTS | 27 |
| | 6.1. | Inve | stigational Product and Other Study Treatment | 27 |
| | 6.2. | Med | ical Device | 28 |
| | 6.3. | Trea | tment Assignment | 28 |
| | 6.4. | Adm | ninistration Schedule (Starting Dose, Dose Adjustment, and | |
| | | Dosi | ing Frequency) | 29 |
| | 6.4 | l.1. | Daprodustat | 29 |
| | 6 | 6.4.1.1. | Starting Dose | 29 |
| | 6 | 6.4.1.2. | Maintenance Dose | 29 |
| | 6.4 | l.2. | Darbepoetin Alfa | 30 |
| | 6 | 6.4.2.1. | Dose Conversion | 30 |
| | 6 | 6.4.2.2. | Maintenance Dose | 31 |

| | 6.5. | Blin | ding | 31 |
|---|---|---|---|---|
| | 6.6. | Pacl | kaging and Labeling | 32 |
| | 6.7. | Prep | paration/Handling/Storage/Accountability | 32 |
| | 6.8. | Con | pliance with Study Treatment Administration | 33 |
| | 6.9. | Trea | tment of Study Treatment Overdose | 33 |
| | 6.10. | Trea | tment after the End of the Study | 34 |
| | 6.11. | Con | comitant Medications and Non-Drug Therapies | 34 |
| | 6.11. | .1. | Permitted Medications and Non-Drug Therapies | 34 |
| | 6.11. | .2. | Prohibited Medications and Non-Drug Therapies | 34 |
| | 6.12. | Sup | plemental Iron Therapy | 34 |
| 7 | . Stud | ly As | sessments and Procedures | 35 |
| | 7.1. | Time | and Events Table | 35 |
| | 7.2. | Scre | ening and Critical Baseline Assessments | 39 |
| | 7.3. | Effic | асу | 39 |
| | 7.4. | Safe | ty | 39 |
| | 7.4.1 | | Adverse Events (AE) and Serious Adverse Events (SAEs) | 39 |
| | 7.4 | 4.1.1. | Time period and Frequency for collecting AE and SAE information | 39 |
| | 7.4 | 4.1.2. | Method of Detecting AEs and SAEs | 40 |
| | 7.4 | 4.1.3. | Follow-up of AEs and SAEs | 40 |
| | 7.4 | 4.1.4. | Cardiovascular and Death Events | 40 |
| | 7.4 | 4.1.5. | Regulatory Reporting Requirements for SAEs | 41 |
| | 7.4.2 | <u>).</u> | Adverse Events of Special Interest | 41 |
| | 7.4.3 | 3. | Pregnancy | 41 |
| | 7.4.4 | J. | Medical Device Incidents (Including Malfunctions) | 42 |
| | 7.4 | 4.4.1. | Time Period for Detecting Medical Device Incidents | 42 |
| | 7.4 | 4.4.2. | Follow-up of Medical Device Incidents | 42 |
| | 7.4 | 4.4.3. | Prompt Reporting of Medical Device Incidents to GSK | 42 |
| | 7.4.5 | j. | Vital Signs/Height/Weight | 43 |
| | 7.4.6 | <b>)</b> . | Electrocardiogram (ECG) | 43 |
| | 7.4.7 | <b>'</b> . | Clinical Laboratory Assessments | 43 |
| | 7.4.8 | <b>3.</b> | Ophthalmology | 44 |
| | 7.5. | Pha | rmacokinetics | 44 |
| | 7.6. | Gen | etics | 45 |
| | 7.7. | Pati | ent Reported Outcome (PRO) | 45 |
| | 7.7.1 | ١. | Health Related Quality of Life (SF-36) | 45 |

| | 7.7.2 | 2. EuroQol 5 Dimension 5 Level Health Utility Index (EQ-5D-5L)/ EuroQol Visual Analogue Scale (EQ-VAS) | 45 |
|---|---|---|---|
| 8. | DAT | A MANAGEMENT | |
| 9. | | TISTICAL CONSIDERATIONS AND DATA ANALYSES | |
| , | 9.1. | Hypotheses | |
| , | 9.2. | Sample Size Considerations | 47 |
| | 9.2. | · | |
| | 9.2.2 | 2. Sample Size Sensitivity | 47 |
| | 9.2. | 3. Sample Size Re-estimation or Adjustment | 47 |
| , | 9.3. | Data Analysis Considerations | |
| | 9.3. | 1. Analysis Populations | 47 |
| | 9.3.2 | 2. Interim Analysis | 48 |
| | 9.3. | 3. Adjustment for Multiplicity | 48 |
| , | 9.4. | Key Elements of Analysis Plan | 48 |
| | 9.4. | 1. Primary Efficacy Analysis | 48 |
| | 9.4.2 | 2. Principal Secondary Efficacy Analysis | 49 |
| | 9.4. | 3. Other Secondary Efficacy Analyses | 49 |
| | 9.4.4 | 4. Safety Analyses | 49 |
| | 9. | 4.4.1. Exposure | 50 |
| | 9. | 4.4.2. Adverse Events | 50 |
| | 9. | 4.4.3. Other Safety Parameters | 50 |
| | 9.4. | 5. Pharmacokinetics Analyses | 50 |
| | 9.4.0 | 6. PRO Data Analysis | 50 |
| 10 | . STU | DY GOVERNANCE CONSIDERATIONS | 51 |
| | 10.1. | Posting of Information on Publicly Available Clinical Trial Registers | 51 |
| | 10.2. | Regulatory and Ethical Considerations, Including the Informed | |
| | | Consent Process | |
| | 10.3. | Quality Control (Study Monitoring) | |
| | 10.4. | Quality Assurance | |
| | 10.5. | Study and Site Closure | |
| | 10.6. | Records Retention | 53 |
| | 10.7. | Provision of Study Results to Investigators, Posting of Information | |
| | 40.0 | on Publically Available Clinical Trials Registers and Publicatio | |
| | 10.8. | Study Period | |
| | 10.9.<br>DEE | Study Administrative Structure | |
| | | ERENCES | |
| ı۷ | . APP | PENDICES | อต |

| 12.1. | App | endix 1: Abbreviations and Trademarks | .56 |
|---|---|---|---|
| 12.2. | App | endix 2: Risk Assessment | .58 |
| 12.3. | Appe | endix 3: Modified List of Highly Effective Methods for Avoiding | |
| | Preg | nancy in Females of reproductive potential | .64 |
| 12.4. | App | endix 4: Collection of Pregnancy Information | .65 |
| 12.5. | Appe | endix 5: Liver Safety Required Actions and Follow up | |
| | Asse | essments | .66 |
| 12.6. | Appe | endix 6: Definition of and Procedures for Recording, Evaluating, | |
| | Follo | ow-Up and Reporting of Adverse Events | .69 |
| 12.6 | .1. | Definition of Adverse Events | .69 |
| 12.6 | .2. | Definition of Serious Adverse Events | .70 |
| 12.6 | .3. | Definition of Cardiovascular Events | .71 |
| 12.6 | .4. | Recording of AEs and SAEs | .71 |
| 12.6 | .5. | Evaluating AEs and SAEs | .72 |
| 12.6 | .6. | Reporting of SAEs to GSK | |
| 12.7. | Appe | endix 7 - Genetic Research | |
| 12.8. | | endix 8: Definition of and Procedures for Documenting Medical | |
| 12.0. | | ce Incidents we are a recording for Bocumenting Medical | .77 |
| 12.8. | | Definitions of a Medical Device Incident | |
| 12 | 2.8.1.1 | | |
| 12.9. | App | endix 9: Protocol Changes | .79 |
| 12.9. | .1. | Amendment 1 — Summary of Changes and Rationale | .79 |
| 12.9 | .2. | Amendment 2 — Summary of Changes and Rationale | .82 |

# 1. PROTOCOL SYNOPSIS FOR STUDY PHI201754

# Rationale

This Phase III study will evaluate the efficacy and safety of daprodustat following a switch from erythropoietin-stimulating agents (ESA) in Japanese subjects with anemia associated with chronic kidney disease (CKD) on hemodialysis (HD) who are currently treated with ESA. The primary objective is to demonstrate non-inferiority of daprodustat to darbepoetin alfa based on hemoglobin (Hgb) in the HD patient population included in this study. Study results will be used as pivotal study data for an NDA submitted for daprodustat for the treatment of renal anemia in Japan.

# Objective(s)/Endpoint(s)

| Objective | Endpoint |
|---|---|
| Primary (efficacy) | |
| To demonstrate non-inferiority of<br>daprodustat to darbepoetin alfa based on<br>hemoglobin (Hgb) | Mean Hgb during the primary efficacy<br>evaluation period (Weeks 40 to 52) |
| Principal secondary (efficacy) | |
| To demonstrate superiority of daprodustat<br>to darbepoetin alfa in terms of<br>achievement/maintenance of target Hgb | Number (%) of subjects with mean Hgb in the target range (10.0-12.0 g/dL) during the primary efficacy evaluation period (Weeks 40 to 52) |
| Other secondary (efficacy, PK) | |
| To evaluate the appropriateness of the starting dose of daprodustat | <ul> <li>Change from baseline in Hgb at Week 4 (Hgb increase rate)</li> <li>Number (%) of subjects by Hgb change from baseline category at Week 4</li> </ul> |
| To evaluate dose adjustment scheme of daprodustat | <ul> <li>Distribution of the dose level</li> <li>Duration of treatment interruption due to Hgb &gt;13.0 g/dL</li> <li>Frequency of dose adjustments</li> </ul> |
| To evaluate the overall Hgb control of daprodustat using darbepoetin alfa as control | <ul> <li>Hgb and change from baseline at each assessment visit</li> <li>Number (%) of subjects who have a Hgb level within the target range (10.0–12.0 g/dL) at each assessment visit</li> <li>Time (%) in Hgb target range (10.0–12.0 g/dL) during the primary efficacy evaluation period (Weeks 40 to 52)</li> <li>Number (%) of subjects who have an Hgb level of less than 7.5 g/dL</li> <li>Number (%) of subjects who have an Hgb increase of more than 2.0 g/dL over any 4</li> </ul> |

| Objective | Endpoint |
|---|---|
| | <ul> <li>weeks</li> <li>Number (%) of subjects who have an Hgb level of more than 13.0 g/dL and number of episodes</li> </ul> |
| To evaluate the PK of daprodustat | AUC and Cmax of plasma daprodustat |
| Exploratory | |
| To evaluate the effect of daprodustat on iron use using darbepoetin alfa as control | <ul> <li>Dose of i.v. iron during the study period and the primary efficacy evaluation period (Weeks 40 to 52)</li> <li>Number (%) of subjects who use i.v. iron during the study period and the primary efficacy evaluation period (Weeks 40 to 52)</li> </ul> |
| To evaluate the effect of daprodustat on iron metabolism using darbepoetin alfa as control | <ul> <li>Change from baseline in ferritin</li> <li>Change from baseline in transferrin saturation (TSAT)</li> <li>Changes from baseline in hepcidin</li> <li>Change from baseline in serum iron</li> <li>Change from baseline in total iron binding capacity (TIBC)</li> </ul> |
| Patient reported outcome | |
| To evaluate the effect of daprodustat on<br>health-related QoL (HR-QoL) using<br>darbepoetin alfa as control | <ul> <li>SF-36</li> <li>Changes from baseline in SF-36 HRQoL scores [Physical Component Summary (PCS), Mental Component Summary (MCS), and 8 subscales] at Week 12, 28 and 52</li> <li>EQ-5D-5L/EQ-VAS</li> <li>Change from baseline in EQ-5D-5L score at Week 12, 28 and 52</li> <li>Change from baseline in EQ-VAS at Week 12, 28 and 52</li> </ul> |
| Safety | 1 |
| To evaluate the safety and tolerability of<br>daprodustat using darbepoetin alfa as<br>control | <ul> <li>Incidence and severity of AEs and SAEs, including AEs of special interest</li> <li>Reasons for discontinuation of study medication</li> <li>Laboratory tests, ECG, vital signs, and ophthalmology assessments</li> </ul> |

## **Study Design**

This is a Phase III, double-blind (double-dummy), active-controlled, parallel-group, multi-center study designed to evaluate the efficacy (non-inferiority) and safety of daprodustat, when administered for 52 weeks, compared to darbepoetin alfa in approximately 270 Japanese HD subjects with anemia associated with CKD who are currently treated with ESA.

Approximately 270 eligible HD subjects will be randomized in a 1:1 ratio on Day 1to receive daprodustat or darbepoetin alfa (approximately 135 subjects per group).

This study consists of a 2~4 week screening phase, a 52 week treatment phase [including the primary efficacy evaluation period (Weeks 40 to 52)], and a 2-week follow-up phase following the treatment phase. The study design is shown below.



# Method of Administration of Study Medication in Each Treatment Group

In each treatment group, study medication will be administered as follows:

- Daprodustat group: Subjects will receive oral daprodustat once daily and intravenous darbepoetin alfa matching placebo once weekly. Daprodustat will be started at a dose of 4 mg once daily (starting dose) on Day 1. From Week 4 onwards, dose adjustments will be made within the dose range of 1-24 mg every 4 weeks according to the prespecified dose adjustment algorithm to achieve and/or maintain Hgb within the target range (10.0-12.0 g/dL).
- Darbepoetin alfa group: Subjects will receive oral daprodustat matching placebo once daily and intravenous darbepoetin alfa once weekly. Prior ESA therapy will be replaced with intravenous treatment with darbepoetin alfa at the corresponding dose once weekly according to the prespecified dose conversion. Subsequently, dose adjustments will be made within the dose range of 10-60 μg once every 2 weeks according to the prespecified dose adjustment algorithm to achieve and/or maintain Hgb within the target range (10.0-12.0 g/dL).

## **Analysis**

Assuming a non-inferiority margin of -1.0 g/dL, a treatment difference of 0.0 g/dL, and a standard deviation of 1.5 g/dL for mean Hgb during the primary efficacy evaluation period in HD subjects, two-sample t-test has at least 99% power at a one-sided significance level of 2.5% (i.e. two-sided

significance level of 5%) with a sample size of 100 subjects per group. Assuming a dropout rate of approximately 25%, approximately 135 subjects will be randomized to each group.

The primary endpoint, which is the mean Hgb during the primary efficacy evaluation period, will be analyzed to demonstrate the non-inferiority of daprodustat to darbepoetin alfa in HD subjects. A mixed model for repeated measurements (MMRM) will be used to estimate the mean Hgb during the primary efficacy evaluation period and its 95% CI by treatment groups. As a preliminary assessment, it will be confirmed if the lower and upper limit of 95% CI for mean Hgb during the primary efficacy evaluation period in daprodustat group would lie fully within target range (10.0-12.0 g/dL) at first. In addition, the point estimate and 95% CI for the treatment difference (daprodustat - darbepoetin alfa) in mean Hgb during the primary efficacy evaluation period will be estimated. Non-inferiority will be established if the lower limit of the 95% CI is greater than -1.0 g/dL. Even if the 95% CI for the difference is completely negative (i.e. lies fully within the range -0.75 to <0 g/dL) non-inferiority would still be concluded on condition that the mean Hgb estimate in the daprodustat group is within the target range.

The primary efficacy population will be the Intent-to-Treat (ITT) Population, and the analysis will be repeated in the modified ITT (mITT) and Per-Protocol (PP) Population to evaluate the robustness of the conclusion. Following sensitivity analyses will be conducted to assess robustness of study result.

- If there are Hgb considered to be impacted by blood transfusion or marketed rhEPO/ESAs, sensitivity analysis excluding the Hgb values from the analyses of primary endpoint will be conducted.
- Analysis of covariance (ANCOVA) will be conducted as sensitivity analysis to MMRM. This model includes treatment group and baseline Hgb. The analysis population will be mITT population and the similar analysis will be repeated in the PP population.
- A tipping point analysis based on multiple imputation will be conducted as sensitivity analysis to
  missing data assumption. This analysis explores a point where non-inferiority is not confirmed
  (tipping point) by changing assumption to missing data and repeating imputation. The analysis
  population will be ITT population and the similar analysis will be repeated in the mITT and PP
  population.

Further details of sensitivity analyses will be provided in the Reporting and Analysis Plan (RAP).

The principal secondary endpoint, which is the proportion of subjects whose mean Hgb during the primary efficacy evaluation period is within the target range, will be analyzed to demonstrate the superiority of daprodustat to darbepoetin alfa in HD subjects.

In the mITT Population, a logistic regression model including treatment group and baseline Hgb as covariates will be used to estimate the point estimate and 95% CI for the odds ratio (daprodustat / darbepoetin alfa). This analysis will be performed to demonstrate the superiority at a two-sided significance level of 5%, conditional on the primary endpoint achieving noninferiority. Superiority will be established if the lower limit of the 95% CI for the odds ratio is greater than 1.0.

#### 2. INTRODUCTION

Daprodustat is a hypoxia-inducible factor (HIF)-prolyl hydroxylase inhibitor (PHI) that stimulates erythropoiesis in the same manner as innate response to hypoxia and is currently being developed as a new treatment for renal anemia.

## 2.1. Study Rationale

This is a Phase III study to evaluate the efficacy and safety of daprodustat following a switch from ESA in Japanese HD subjects with renal anemia who are currently treated with ESA. The primary objective is to demonstrate non-inferiority of daprodustat to darbepoetin alfa based on Hgb in the HD patient population included in this study. Study results will be used as pivotal study data for an NDA submitted for daprodustat for the treatment of renal anemia in Japan.

## 2.2. Background

Renal anemia is diagnosed in many patients with CKD, and the prevalence of renal anemia increases with progression of CKD [Akizawa, 2011]. Causes of anemia in CKD patients include absolute or relative deficiency of erythropoietin (EPO), shortened erythrocyte survival, and reduced iron availability. Anemia is further exacerbated by chronic blood loss associated with hemodialysis procedure, infection, and functional hemolysis [Japanese Society for Dialysis Therapy, 2016].

Daprodustat is a hypoxia-inducible factor-prolyl hydroxylase inhibitor that is currently being developed as a treatment for renal anemia. Data in Japanese patients have been collected from a Japanese Phase II 4-week treatment study in Japanese hemodialysis (HD) subjects (PHI116099: 97 Japanese subjects), an international multi-center Late Phase II 24-week treatment study in HD subjects (PHI113633: including 24 Japanese subjects), and an international multi-center Late Phase II 24-week treatment study in Non-dialysis subjects (PHI113747: including 42 Japanese subjects). In these clinical studies, daprodustat increased endogenous EPO, reduced hepcidin, and increased Hgb in HD and ND subjects including Japanese subjects. In addition, daprodustat increased Hgb at lower blood EPO concentrations than existing ESAs.

Summaries of findings from both clinical and non-clinical studies conducted with daprodustat can be found in the daprodustat Investigator's Brochure (IB) and IB supplement(s) (if applicable). A benefit: risk assessment, including risk mitigation strategies, is outlined in Section 4.6.

# 3. OBJECTIVES AND ENDPOINTS

| | Objective | Endpoint |
|---|---|---|
| Pri | mary (efficacy) | |
| • | To demonstrate non-inferiority of<br>daprodustat to darbepoetin alfa based on<br>hemoglobin (Hgb) | Mean Hgb during the primary efficacy<br>evaluation period (Weeks 40 to 52) |
| Pri | ncipal secondary (efficacy) | , |
| • Otl | To demonstrate superiority of daprodustat to darbepoetin alfa in terms of achievement/maintenance of target Hgb her secondary (efficacy, PK) | Number (%) of subjects with mean Hgb in the target range (10.0-12.0 g/dL) during the primary efficacy evaluation period (Weeks 40 to 52) |
| • | To evaluate the appropriateness of the starting dose of daprodustat | <ul> <li>Change from baseline in Hgb at Week 4 (Hgb increase rate)</li> <li>Number (%) of subjects by Hgb change from baseline category at Week 4</li> </ul> |
| • | To evaluate dose adjustment scheme of daprodustat | <ul> <li>Distribution of the dose level</li> <li>Duration of treatment interruption due to Hgb &gt;13 g/dL</li> <li>Frequency of dose adjustments</li> </ul> |
| • | To evaluate the overall Hgb control of daprodustat using darbepoetin alfa as control | <ul> <li>Hgb and change from baseline at each assessment visit</li> <li>Number (%) of subjects who have a Hgb level within the target range (10.0–12.0 g/dL) at each assessment visit</li> <li>Time (%) in Hgb target range (10.0–12.0 g/dL) during the primary efficacy evaluation period (Weeks 40 to 52)</li> <li>Number (%) of subjects who have an Hgb level of less than 7.5 g/dL</li> <li>Number (%) of subjects who have an Hgb increase of more than 2 g/dL over any 4 weeks</li> <li>Number (%) of subjects who have an Hgb level of more than 13.0 g/dL and number of episodes</li> </ul> |
| • | To evaluate the PK of daprodustat | AUC and Cmax of plasma daprodustat |
| Ex | ploratory | |
| • | To evaluate the effect of daprodustat on iron use using darbepoetin alfa as control | <ul> <li>Dose of i.v. iron during the study period and the primary efficacy evaluation period (Weeks 40 to 52)</li> <li>Number (%) of subjects who use i.v. iron during the study period and the primary</li> </ul> |

| Objective | Endpoint |
|---|---|
| | efficacy evaluation period (Weeks 40 to 52) |
| To evaluate the effect of daprodustat on | Change from baseline in ferritin |
| iron metabolism using darbepoetin alfa control | Change from baseline in transferrin saturation (TSAT) |
| | Changes from baseline in hepcidin |
| | Change from baseline in serum iron |
| | • Change from baseline in total iron binding capacity (TIBC) |
| Patient reported outcome | |
| To evaluate the effect of daprodustat on | SF-36 |
| health-related QoL (HR-QoL) using darbepoetin alfa as control | • Changes from baseline in SF-36 HR-QoL scores [Physical Component Summary (PCS), |
| | Mental Component Summary (MCS), and 8 subscales] at Week 12, 28 and 52 |
| | EQ-5D-5L/ EQ-VAS |
| | <ul> <li>Change from baseline in EQ-5D-5L score at<br/>Week 12, 28 and 52</li> </ul> |
| | • Change from baseline in EQ-VAS at Week 12, 28 and 52 |
| Safety | , |
| To evaluate the safety and tolerability of daprodustat using darbepoetin alfa as | including AEs of special interest |
| control | Reasons for discontinuation of study medication |
| | • Laboratory tests, ECG, vital signs, and ophthalmology assessments |

CONFIDENTIAL

#### 4. STUDY DESIGN

## 4.1. Overall Design

This is a Phase III, double-blind (double-dummy), active-controlled, parallel-group, multi-center study designed to evaluate the efficacy (non-inferiority) and safety of daprodustat, when administered for 52 weeks, compared to darbepoetin alfa in approximately 270 Japanese HD subjects with anemia associated with CKD who are currently treated with ESA.

Two hundreds seventy (270) eligible HD subjects will be randomized in a 1:1 ratio to receive daprodustat or darbepoetin alfa (135 subjects per group).

This study consists of a 2~4 week screening phase, a 52 week treatment phase [including the primary efficacy evaluation period (Weeks 40 to 52)], and a 2-week follow-up phase following the treatment phase. The study design is shown in Figure 1.



# 4.2. Treatment Groups and Study Periods

Details for each study period and treatments are described below. In this study, a point-of-care Hgb analyzer (HemoCue®) will consistently be utilized for confirmation of subjects' eligibility, withdrawal criteria and dose adjustments of study medication.

#### Screening phase

Subjects who have provided informed consent and meet all of the eligibility criteria at screening (Week -4~-2) (Sections 5.1 and 5.2) will be provisionally enrolled in the study. Subjects who have used oral iron since before the start of the study must remain on the same regimen throughout the screening phase (intravenous iron will not be allowed). Subjects will also continue to use ESA throughout the screening phase. The regimen of ESA therapy should remain unchanged throughout the screening phase.

## **Treatment phase**

Subjects who meet all of the eligibility criteria at the start of the treatment phase (Day 1) will be randomized in a 1:1 ratio to receive daprodustat or darbepoetin alfa and enrolled in the study. Subjects will be ESA users and will switch their ESA therapy to darprodustat at Day 1 so that the randomization date (Day 1) should coincide, as closely as possible, with the date of next scheduled ESA administration. In accordance with the randomization instructions, subjects randomized to the daprodustat group will receive daprodustat and darbepoetin alfa matching placebo for 52 weeks. Subjects randomized to the darbepoetin alfa group will receive daprodustat matching placebo and darbepoetin alfa for 52 weeks. Daprodustat will be orally administered once daily, and darbepoetin alfa will be intravenously administered once weekly. In both groups, dose adjustments for study medication during the treatment phase will be made according to the administration schedule specified in Section 6.4 to achieve and/or maintain Hgb within the target range (10.0-12.0 g/dL). In addition, supplemental iron therapy will be administered according to the standard initiation criteria as described in Section 6.12. It should be noted that intravenous iron or dose change for oral iron will not be allowed from Day 1 to Week 4.

## Follow-up phase

Subjects will visit the site for follow-up assessments and observations 2 weeks after the completion/discontinuation of study treatment. During the follow-up phase, treatment of renal anemia will be allowed as necessary at the discretion of the investigator (or subinvestigator).

## 4.3. Study Subjects and Number of Subjects

A total of 270 subjects will be randomized (daprodustat group: 135 subjects, darbepoetin alfa group: 135 subjects). Assuming a dropout rate of 30% during the screening phase, approximately 386 subjects need to be screened. Assuming a dropout rate of 25% after the start of study treatment, a total of 202 subjects are expected to complete the 52-week treatment.

Table 1 Target Number of Subjects

| Screened | 386 |
|-----------------------------|-----|
| Randomized/enrolled | 270 |
| Completed 52-week treatment | 202 |

# 4.4. Rationale for Study Design

#### **Objectives and evaluations**

This is a Phase III study to evaluate the efficacy and safety of daprodustat in Japanese HD subjects with renal anemia who are currently treated with ESA. The study is designed as an active-controlled, parallel-group comparative study which will be conducted under double blind to meet the primary objective, that is, to demonstrate non-inferiority of daprodustat to the existing drug based on Hgb in HD subjects. The target Hgb range was set for study treatment in line with the Guidelines for Renal Anemia in Chronic Kidney Disease issued by the Japanese Society for Dialysis Therapy in 2015 [The Japanese Society for Dialysis Therapy, 2016] to demonstrate that treatment with daprodustat can

result in achievement and/or maintenance of target Hgb in HD subjects, and evaluate the appropriateness of the starting dose of daprodustat.

## Control

Darbepoetin alfa, which has been widely used in Japanese patients with renal anemia, primarily HD patients, since its approval in Japan in 2007, was selected as control.

#### 4.5. Rationale for Dose Levels

## Starting dose and dose adjustments of daprodustat

The starting dose (4 mg) and the dose adjustment method (maintenance dose range: 1-24 mg) for daprodustat are described in Section 6.4.

The starting dose and the dose adjustment algorithm selected for Japanese HD subjects in the present study are based on the results from a review of the longitudinal model constructed using Hgb data from six Japanese or overseas Phase II studies (PHI112844, PHI116581, PHI116582, PHI113633, PHI113747, and PHI116099) as well as the results from clinical studies. The data set used in the model analyses was based on the data of daprodustat administered in a wide dose range (0-25 mg) and included a Japanese Phase II 4-week treatment study (PHI116099) and international multi-center late Phase II 24-week treatment studies (PHI113633 and PHI113747) in which subjects in Japan participated.

## Starting dose

Simulations using a longitudinal model as well as clinical data for HD subjects suggested that Hgb levels observed with prior ESA therapy is maintained for 4 weeks after a switch from prior ESA to study medication, with no rapid increase greater than 2 g/dL, at the dose level of 4 mg in ESA user subjects. Covariate analyses identified baseline Hgb, body weight, and dose level of prior ESA as major factors affecting Hgb. However, Hgb was more greatly affected by inter-subject differences in drug response to daprodustat than these factors.

Taken together, 4 mg may be an appropriate starting dose of daprodustat for the majority of ESA users.

#### Maintenance dose range and dose adjustment algorithm

Simulation results using the longitudinal model showed that drug response to daprodustat regarding Hg greatly varied among subjects, indicating that the dose range from 1 to 24 mg may be necessary to achieve and maintain target Hgb. Accordingly, a total of 8 dose levels (1, 2, 4, 6, 8, 12, 18, and 24 mg) were selected as the maintenance doses, with 4 mg intended for subjects with a standard drug response. The dose adjustment algorithm was defined so that target Hgb (10.0-12.0 g/dL) set for the present study according to the Guidelines for Renal Anemia [The Japanese Society for Dialysis Therapy, 2016] can be maintained. Given a difference of 1.0 g/dL between the the upper limit of Hgb target range (12.0 g/dL) and ESA dose interruption criteria value (13.0 g/dL), the dose of daprodustat will be reduced to the one step lower dose level when Hgb increases into the range of 12.0−13.0 g/dL. Since it is well known that an Hgb increase of 0.5 g/dL or less per week is appropriate to prevent adverse reactions, the dose level will be reduced by one step when Hgb increases by more than 2 g/dL over 4 weeks [KDIGO, 2012]. For subjects whose anemia needs to be corrected (≥7.5 g/dL and <10.0 g/dL),

the dose level will be maintained while the Hgb increase per 4 weeks is 0.5-2 g/dL, and the dose level will be increased by one step when the Hgb increase per 4 weeks is less than 0.5 g/dL.

# Starting dose and dose adjustments of control (darbepoetin alfa)

The starting doses and dose adjustment algorithm for darbepoetin alfa are described in Section 6.4. The starting doses of darbepoetin alfa for subjects currently treated with epoetin were selected based on the prescribing information in Japan. For subjects on epoetin beta pegol, given that no recommended starting doses of darbepoetin alfa when switched from epoetin beta pegol approved in Japan is available, switchig will be performed in the epoetin beta pegol-to-darbepoetin alfa dose ratio of 5:6 at the middle dose level of darbepoetin alfa according to the overseas prescribing information [MIRCERA. Product information in Europe, 2012]. At the other dose levels, dose conversion will be performed within the approved dose levels and in a dose ratio close to 5:6.

The dose adjustment algorithm for darbepoetin alfa was determined based on the product information and previous Japanese clinical studies in accordance with the Guideline for Renal Anemia in Chronic Kidney Disease [Japanese Association for Dialysis Therapy, 2016].

#### 4.6. Benefit: Risk Assessment

Summaries of findings from clinical and nonclinical studies of daprodustat can be found in the IB and the IB supplements. The risk assessment and risk minimization strategies for the present study are outlined in the following sections:

#### 4.6.1. Risk Assessment

The potential risks of clinical significance including AEs of special interest (Section 7.4.2) and the mitigation strategies for this protocol taking into account the results of completed clinical and nonclinical studies of daprodustat, are outlined in Section 12.2. Appendix 2.

#### 4.6.2. Benefit Assessment

Study PHI201754 is a Phase 3 study in Japanese HD subjects with renal anemia who are treated with ESA. Previous clinical studies of daprodustat, administered for up to 24 weeks in ND or HD subjects have demonstrated clinical efficacy (increase in and/or maintenance of Hgb) with blood EPO concentrations increased within the normal physiologic range in CKD subjects. Data obtained in Study PHI201754 will generate safety and efficacy data in Japanese HD subjects with renal anemia who are treated with ESA, for a 52-week treatment period. Study participants who will receive daprodustat, may benefit from the expected clinical efficacy.

Daprodustat, may have important advantages over existing ESAs. Daprodustat, which is orally administered and requires no cold chain management unlike ESAs, is more convenient to patients and health care provider. Daprodustat is shown to increase Hgb at lower EPO concentrations than ESAs. Since increased exposure to EPO following administration of ESAs may be associated with an increased cardiovascular risk [Szczech, 2008], daprodustat may increase Hgb without increasing the cardiovascular risk.

## 4.6.3. Overall Benefit: Risk Conclusion

Daprodustat is shown to have a positive benefit-risk balance based on the following findings: in studies of daprodustat administered for up to 24 weeks, treatment with daprodustat resulted in achievement of target Hgb, and no adverse events have been identified as related to treatment with daprodustat.

This protocol employs precautions to mitigate known and potential risks to enrolled subjects (see Section 12.2. Appendix 2). Given these precautions, as well as the potential benefit that daprodustat holds for the treatment of renal anemia compared with the current standard treatment, the overall benefit risk balance is considered to be positive.

#### 5. SUBJECT SELECTION AND WITHDRAWAL CRITERIA

Specific information regarding warnings, precautions, contraindications, adverse events, and other pertinent information on the GSK investigational product or other study treatment that may impact subject eligibility is provided in the IB/IB supplement(s) and/or other pertinent documents.

Deviations from inclusion/exclusion criteria are not allowed because they can potentially jeopardize the scientific integrity of the study, regulatory acceptability or subject safety. Therefore, adherence to the criteria as specified in the protocol is essential.

#### 5.1. Inclusion Criteria

Subjects eligible for enrolment in the study must meet all of the inclusion criteria.

Note: Verification at both provisional enrolment (screening) and official enrolment (Day 1) is required, unless otherwise specified.

- 1. Age (informed consent): ≥20 years of age
- 2. Dialysis: On hemodialysis (HD) or hemodiafiltration (HDF) given three times weekly for at least 12 weeks prior to screening
- 3. ESAs: Use of one and the same ESA for at least 10 weeks prior to screening
- 4. ESA dose: Darbepoetin alfa 10 60 µg per week, epoetin (including biosimilars) ≤9000 IU per week, or epoetin beta pegol up to 250 µg per 4 weeks Note: ESA dose must be greater than the minimum ESA dose if Hgb >12 g/dL to 12.5 g/dL (Minimum ESA dose: epoetins (including biosimilars): 1500 units (U) per week; darbepoetin alfa: 10 µg per week; epoetin beta pegol: 25 µg per evey 4 weeks)
- 5. Hemoglobin (Hgb): ≥9.5 g/dL and ≤12.5 g/dL. Determined at the site using an Hgb analyzer (HemoCue®)
- 6. Iron parameters: Ferritin > 100 ng/mL or TSAT > 20% (screening verification only)
- 7. Gender (screening verification only): Female or male
  Females: Not pregnant [demonstrated to be negative for human chorionic gonadotropin (hCG) in
  serum], not breast-feeding, and meet at least one of the following:
  - 1) Females of non-childbearing potential are defined as follows:
  - Pre-menopausal with at least one of the following and no plans to utilise assisted reproductive techniques (e.g., in vitro fertilisation or donor embryo transfer):
    - History of bilateral tubal ligation or salpingectomy
    - History of hysteroscopic tubal occlusion and postoperatively documented bilateral tubal obstruction
    - History of hysterectomy
    - History of bilateral oophorectomy
  - Postmenopausal defined as A) females 60 years of age or older or B) In females < 60 years of age, 12 months of spontaneous amenorrhea [in questionable cases a blood sample with postmenopausal follicle stimulating hormone (FSH) and estradiol concentrations is confirmatory (see separately specified reference ranges)]. Females on HRT whose menopausal status is in doubt will be required to use one of the most effective contraception

- methods if they wish to continue their HRT during the study. Otherwise they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
- 2) Females of childbearing potential must agree to comply with one of the contraception methods listed as requirements in "GSK Listing of Most Effective Contraceptive Methods for Females of Childbearing Potential (Section 12.3. Appendix 3: Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of reproductive potential)" from at least 28 days prior to the first dose of study medication until the completion of the follow-up visit.
- 8. Informed consent: Written informed consent, including adherence to the requirements and conditions specified in the consent form and the protocol, must be obtained from each subject as specified in Section10.2...

#### 5.2. Exclusion Criteria

Subjects meeting any of the following criteria must not be enrolled in the study.

Note: Verification at both provisional enrolment (screening) and official enrolment (Day 1) is required, unless otherwise specified.

# Chronic kidney disease (CKD)-related criteria

1. Kidney transplant: Planned living-related kidney transplant during the study

#### Anemia-related criteria

- 2. Aplasia: History of bone-marrow hypoplasia or pure red cell aplasia
- 3. Other causes of anemia: pernicious anemia, thalassemia, sickle cell anemia, or myelodysplastic syndromes
- 4. Gastrointestinal (GI) bleeding: Evidence of actively bleeding gastric, duodenal, or esophageal ulcer disease OR clinically significant GI bleeding within 10 weeks prior to screening or during a period from screening to Day 1.

#### Cardiovascular disease-related criteria

- 5. Myocardial infarction, acute coronary syndrome, stroke, or transient ischemic attack: Diagnosed within 10 weeks prior to screening or during a period from screening to Day 1.
- 6. Heart failure: Chronic Class IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system
- Corrected QT (QTc) Interval (screening verification only): QTc >500 msec; or QTc >530 msec in subjects with bundle branch block

Note: <u>QT interval corrected using the Bazett's formula (QTcB)</u> will be used, and ECG can be mechanically or manually read.

#### Other disease-related criteria

- 8. Liver disease (if any of the following occurs):
  - (Screening verification only): Alanine transaminase (ALT) >2×upper limit of normal (ULN)
  - (Screening verification only): Bilirubin >1.5×ULN (isolated bilirubin >1.5×ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%)

 Current unstable active liver or biliary disease (generally defined by the onset of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal/gastric varices, persistent jaundice, or cirrhosis)

CONFIDENTIAL

- Note: Stable liver disease (including asymptomatic gallstones, chronic hepatitis B/C, or Gilbert's syndrome) is acceptable if the subject otherwise meets entry criteria..
- 9. Malignancy: History of malignancy within 2 years prior to screening, currently receiving treatment for cancer, or complex kidney cyst >3 cm (II F, III or IV based on the Bosniak classification)

<u>Note</u>: The only exception is localized squamous cell or basal cell carcinoma of the skin that has been definitively treated  $\geq 10$  weeks before screening.

## Concomitant medication and other study treatment-related criteria

- 10. Iron: Planned use of intravenous iron during the screening phase or during a period from Day 1 to Week 4
  - Note: Oral iron is acceptable. However, the same dose regimen must be used throughout the screening phase and from Day 1 to Week 4. Antihyperphosphatemic agents containing iron (e.g., ferric citrate hydrate) are also acceptable only if used for at least 12 weeks prior to screening. However, they must be continued throughout the screening phase from Day 1 to Week 4.
- 11. Severe allergic reactions: History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product (see the daprodustat IB or the Prescribing Information of the darbepoetin alfa)
- 12. Drugs and supplements: Use or planned use of any prescription or non-prescription drugs or dietary supplements that are prohibited during the study period [prohibited medications: strong inducers and inhibitor of Cytochrome P450 (CYP) 2C8, see Section 6.11.2]
- 13. Prior investigational product exposure: Use of an investigational agent within 30 days or five half lives of the investigational agent (whichever is longer)
- 14. Prior treatment with daprodustat: Any prior treatment with daprodustat for a treatment duration of >30 days

#### General health-related criteria

15. Other conditions: Any other condition, clinical or laboratory abnormality, or examination finding that the investigator (or subinvestigator) considers would put the subject at unacceptable risk, which may affect study compliance or prevent understanding of the aims or investigational procedures or possible consequences of the study

#### 5.3. Screening Failures

Screen failures are defined as subjects who consent to participate in the clinical trial, but are not subsequently randomized in the study. A minimum set of information is required from screen failure subjects including Demography, Screen Failure details, Eligibility Criteria, and SAEs in order to report screen failures in a reliable manner, satisfy the requirements for publication defined by the Consolidated Standards of Reporting Trials (CONSORT), and respond to requests of the regulatory authorities.

Subjects that fail screening are eligible to be rescreened up to 3 times as soon as the investigator assesses they may meet study entry criteria. For re-screening subjects, ophthalmology exam to be performed at re-screening could be replaced with the results of the most recent ophthalmology screening, on the investigator's (or subinvestigator's) discretion (See Table 10).

## 5.4. Permanent discontinuation of study treatment and study withdrawal

If subjects meet one of the following criteria, study treatment should be permanently discontinued and subjects will be withdrawn from the study. The withdrawal reason should be recorded.

- Hgb < 7.5 g/dL
  - Note: HemoCue Hgb values will be employed. If an initial Hgb value meets the Hgb stopping criteria, measurement will be repeated at the same study visit (using the same sample) to calculate the average. If the average meets the Hgb stopping criteria, study treatment will be discontinued.
- Kidney transplant
- Subject becomes pregnant or intends to become pregnant during the study.
- Diagnosis of new or recurrent cancer
- Liver chemistry abnormalities exceeding the threshold criteria (see Section 5.4.1.)
- Need for chronic (more than 14 days) use of prohibited medication (strong inhibitors/ inducers of CYP2C8 meet this criteria)
- When the investigator (or subinvestigator) considers necessary to withdraw the subject from the study for other reasons

Subjects who meet any of the withdrawal criteria or are withdrawn for other reasons during the treatment phase should be assessed at withdrawal visit after study treatment is discontinued, and will then enter the follow-up phase.

Should a subject fail to attend a required study visit, the investigator (or subinvestigator) should take the following measures:

- The investigator (or subinvestigator) or designee should attempt to contact the subject and reschedule the missed visit as soon as possible.
- The investigator (or subinvestigator) should counsel the subject on the importance of maintaining the assigned visit schedule and determine whether the subject is willing to continue his/her participation in the study and/or whether the subject should remain in the study.
- The investigator (or subinvestigator) or designee should make every effort to regain contact with a subject who is deemed "Lost to Follow-up". All efforts to contact the subject should be documented in the subject's clinical charts.
- Should the subject continue to be unreachable, then and only then will he/she be considered "Lost to Follow-up."

A subject may withdraw from the study at any time at his/her own request. The investigator (or subinvestigator) may withdraw a subject from the study at any time for safety or compliance reasons or study conduct considerations. If a subject withdraws from the study, he/she may request destruction

of any clinical samples taken, and the investigator (or subinvestigator) must document this in the site study records.

## 5.4.1. Liver Chemistry Stopping Criteria

**Liver chemistry stopping and increased monitoring criteria** have been designed to assure subject safety and evaluate liver event etiology [in alignment with the Food and Drug Administration (FDA) premarketing clinical liver safety guidance].

## Liver Chemistry Stopping and Increased Monitoring Algorithm



- > Must refer to Liver Safety Required Actions and Follow up Assessments section in the Appendix
- ➤ Report as an SAE if possible Hy's Law case: ALT≥3xULN and Bilirubin≥2xULN (>35% direct) or INR>1.5, if measured\*

\*INR value not applicable to subjects on anticoagulants

# Liver Chemistry Increased Monitoring Algorithm with Continued Therapy for ALT ≥3xULN but <8xULN



Liver Safety Required Actions and Follow up Assessments Section can be found in Section 12.5. Appendix 5

\*INR value not applicable to subjects on anticoagulants

## 5.4.1.1. Study Treatment Restart or Rechallenge

Study treatment restart or rechallenge after liver chemistry stopping criteria are met by any subject participating in this study is not allowed.

## 5.5. Subject and Study Completion

A completed subject is one who has completed all periods of the study including the follow-up visit. The study will be completed with the last subject's last study visit.

#### 6. STUDY TREATMENTS

## 6.1. Investigational Product and Other Study Treatment

The term 'study treatment' is used throughout the protocol to describe any products received by the subject as per the protocol design. Accordingly, 'study treatment' sometimes refers to each product and sometimes refers to multiple products.

## Daprodustat (study drug)

The study drug daprodustat will be supplied as fast-release film coated tablets for oral administration containing 1 mg, 2 mg, 4 mg, or 6 mg of daprodustat (Table 2). The daprodustat matching placebo will be supplied as film coated tablets, it visually matches the daprodustat tablets, for oral administration containing no daprodustat (Table 2). There are two sizes each for the daprodustat and placebo tablets.

Table 2 Description of daprodustat and placebo tablets

| Daprodustat or placebo tablets | Description |
|---|---|
| Daprodustat (small) | 7.0 mm round, standard biconvex, white film coated tablets containing |
| (1 mg, 2 mg, and 4 mg tablets | 1 mg, 2 mg, or 4 mg of daprodustat as active ingredient |
| Daprodustat (large) | 9.0 mm round, standard biconvex, white film coated tablets containing |
| (6 mg tablets) | 6 mg of daprodustat as active ingredient |
| Placebo (small) | 7.0 mm round, standard biconvex, white film coated tablets containing no |
| | daprodustat |
| Placebo (large) | 9.0 mm round, standard biconvex, white film coated tablets containing no |
| | daprodustat |

Daprodustat and placebo tablets are packed by strength or by size in high density polyethylene bottles, with 35 tablets per bottle. Subjects are to take one to four tablets (Table 3) with water once daily according to the dose level indicated at each study visit. Subjects can take daprodustat tablets without regard to food or hemodialysis. The administration schedule (starting dose and dose adjustment) described in Section 6.4.1 should be followed.

Table 3 Dose levels of daprodustat and number of tablets taken

| Dose level of | 1 mg | 2 mg | 4 mg | 6 mg | 8 mg | 12 mg | 18 mg | 24 mg |
|---|---|---|---|---|---|---|---|---|
| daprodustat | | | | | | | | |
| (once daily) | | | | | | | | |
| Number of | 1 mg | 2 mg | 4 mg | 6 mg | 4 mg | 6 mg | 6 mg | 6 mg |
| daprodustat | tablet | tablet | tablet | tablet | tablet | tablet | tablet | tablet |
| tablets taken | $\times 1$ | ×1 | ×1 | ×1 | ×2 | ×2 | ×3 | ×4 |

Subjects should be instructed to bring daprodustat/placebo tablets with bottles at each study visit, and all unused daprodustat tablets will be collected from subjects at every 4 week's study visit.

#### **Darbepoetin Alfa (Control)**

GSK will provide the control drug of darbepoetin alfa (NESP® Injection) and its matching placebo. Darbepoetin alfa is provided as 0.5 mL plastic prefilled syringes (PFS) for IV injection each containing 10, 15, 20, 30, 40 or 60 µg of darbepoetin alfa in a clear and colorless solution.

Darbepoetin alfa placebo is provided as 0.5 mL plastic prefilled syringes (PFS) for IV injection containing no darbepoetin alfa in a clear and colorless solution.

Subjects will receive intravenous darbepoetin alfa or placebo once weekly at the study site (Table 4) according to the dosing schedule (including starting doses and dose adjustment algorithm) provided in Section 6.4.2.

Table 4 Dose levels of darbepoetin alfa and injection frequency

| Dose level of darbepoetin alfa (once weekly) | 10 μg | 15 μg | 20 μg | 30 μg | 40 μg | 60 μg |
|---|---|---|---|---|---|---|
| Number of IV injection of darbepoetin alfa | 10 μg IV | 15 μg IV | 20 μg IV | 30 μg IV | 40 μg IV | 60 μg IV |
| | ×1 | ×1 | ×1 | ×1 | ×1 | ×1 |

#### 6.2. Medical Device

The darbepoetin alfa (Brand name: NESP Injection) marketed with the device (kit formulation which was filled liquid medication in plastic prefilled syringes) provided for use in this study.

Instructions for medical device are described in the Prescribing Information of NESP Injection.

The medical device incidents, including those resulting from malfunctions of the device, must be detected, documented, and reported by the investigator throughout the study – see Section 7.4.4.

## 6.3. Treatment Assignment

The randomization schedule will be generated by GSK statistician using the randomization system (Randall).

Subjects will be randomized centrally in a 1:1 ratio to one of the two treatment groups according to the randomization schedule. Randomization should precede the study treatment.

- Daprodustat group
- Darbepoetin alfa group

Subjects will be assigned a randomization number by the Interactive Web Recognition System (IWRS). Once a randomization number has been assigned, it must not be re-assigned. Further details are provided in the Study Reference Manual (SRM).

# 6.4. Administration Schedule (Starting Dose, Dose Adjustment, and Dosing Frequency)

Instructions regarding container number assignment and dose adjustments for all study treatments are given by the Interactive Web Recognition System (IWRS).

## 6.4.1. Daprodustat

HD subjects randomized to the daprodustat group will receive oral daprodustat according to the following regimen. Furthermore, these subjects will receive i.v. darbepoetin alfa placebo in the same manner with darbepoetin alfa.

## 6.4.1.1. Starting Dose

At Day 1, subjects will skip ESA and will start oral treatment with daprodustat at the starting dose of 4 mg once daily and remain on the same regimen until the day of Week 4.

#### 6.4.1.2. Maintenance Dose

From Weeks 4 to 52, interruption of treatment or dose adjustments will be made within the maintenance dose range of 1-24 mg (Table 5) according to the dose adjustment algorithm (Table 6) to achieve and/or maintain Hgb within the target range (10.0-12.0 g/dL) based on the HemoCue Hgb value measured every 4 weeks. Dose changes will be made every 4 weeks. If any of the one-step dose reduction criteria is met during treatment at the minimum maintenance dose (1 mg), treatment should be interrupted (and administer placebo); once the one-step dose increase criteria are met, treatment at 1 mg will be resumed. If the one-step dose increase criterion is met during treatment at the maximum maintenance dose (24 mg), treatment at 24 mg should be continued.

Table 5 Maintenance dose of daprodustat

| Dose step | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 |
|---|---|---|---|---|---|---|---|---|
| Dose level of | 1 mg | 2 mg | 4 mg | 6 mg | 8 mg | 12 mg | 18 mg | 24 mg |
| daprodustat | | | | | | | | |
| (once daily) | | | | | | | | |
| Number of | 1 mg | 2 mg | 4 mg | 6 mg | 4 mg | 6 mg | 6 mg | 6 mg |
| daprodustat | tablet | tablet | tablet | tablet | tablet | tablet | tablet | tablet |
| tablets taken | $\times 1$ | ×1 | ×1 | ×1 | ×2 | ×2 | ×3 | ×4 |

| | <b>,</b> | , , |
|---|---|---|
| Hgb | Hgb increase over 4 weeks | Treatment |
| (g/dL) | (g/dL) | Treatment |
| >13.0 | NA | Interrupt treatment (and administer placebo) until Hgb decreases to less than 12.0 g/dL, and resume treatment at the one lower dose level [If interrupted (and placebo administered) at 1 mg, |
| | | resume treatment at 1 mg after the one-step dose increase criterion is met] |
| $\geq$ 12.0 and $\leq$ 13.0 | NA | One-step dose reduction |
| ≥10.0 and <12.0 | >2.0 | One-step dose reduction |
| | ≤2.0 | Continue treatment at the current dose level |
| ≥7.5 and <10.0 | >2.0 | One-step dose reduction |
| | 0.5-2.0 | Continue treatment at the current dose level |
| | <0.5 | One-step dose increase |

Table 6 Dose adjustment algorithm (daprodustat)

NA

Discontinue treatment permanently\* and initiate

another appropriate treatment

## 6.4.2. Darbepoetin Alfa

< 7.5

HD subjects randomized to the darbepoetin alfa group will receive intravenous darbepoetin alfa according to the following regimen. Furthermore, these subjects will receive oral daprodustat placebo in the same manner with daprodustat.

#### 6.4.2.1. Dose Conversion

On Day 1, prior ESA will be replaced with darbepoetin alfa at the corresponding dose once weekly (Table 7).

| Table 7 | Replacement with darbepoetin alfa - initial dose (ESA users) |
|---------|--------------------------------------------------------------|
|---------|--------------------------------------------------------------|

| | Prior ESA | |
|---|---|---|
| Epoetin | ≤3000 IU, per week | 15 μg, once weekly |
| | 4500 IU, per week | 20 μg, once weekly |
| | 6000 IU, per week | 30 μg, once weekly |
| | 9000 IU, per week | 40 μg, once weekly |
| Epoetin beta pegol | ≤50 µg, once every 4 weeks* | 15 μg, once weekly |
| | 75 μg, once every 4 weeks* | 20 μg, once weekly |
| | 100 μg, once every 4 weeks* | 30 μg, once weekly |
| | 150 μg, once every 4 weeks* | 40 μg, once weekly |
| | ≥200 µg, once every 4 weeks* | 60 μg, once weekly |
| Darbepoetin alfa | 10, 15, 20, 30, 40, 60 µg, per week | 10, 15, 20, 30, 40, 60 μg, per week |

<sup>\*:</sup> Allowance of ±1 week

Maintenance treatment will be started at Week 2 as described in Section 6.4.2.2.

<sup>\*:</sup> If an initial Hgb value is less than 7.5 g/dL, measurement will be repeated at the same study visit (using the same sample) to calculate the average. If the average meets the Hgb stopping criteria, study treatment will be permanently discontinued.

#### 6.4.2.2. Maintenance Dose

From Weeks 2 to 52, dose interruptions or adjustments will be performed within the maintenance dose range of  $10\sim60~\mu g$  (Table 8) according to the dose adjustment algorithm (Table 9) so that the HemoCue Hgb value measured every other week will achieve or remain within the target range (10.0-12.0 g/dL). Dose adjustments will be made once every 2 weeks. If any of the one-step dose reduction criteria is met during treatment at the minimum maintenance dose ( $10~\mu g$ ), treatment should be interrupted (and placebo administered); once the one-step dose increase criteria are met, treatment at  $10~\mu g$  will be resumed. If the one-step dose increase criterion is met during treatment at the maximum maintenance dose ( $60~\mu g$ ), treatment at  $60~\mu g$  should be continued.

Table 8 Maintenance dose of darbepoetin alfa

| Dose level | 1 | 2 | 3 | 4 | 5 | 6 |
|---|---|---|---|---|---|---|
| Darbepoetin alfa (once weekly) | 10 μg | 15 μg | 20 μg | 30 μg | 40 μg | 60 μg |

Table 9 Dose adjustment algorithm (darbepoetin alfa)

| Hgb (g/dL) | Treatment |
|---|---|
| >13.0 | Interrupt treatment (and administer placebo) until Hgb decreases to less than |
| | 12.0 g/dL, and resume treatment at the one lower dose level |
| | [If interrupted (and placebo administered) at 10 μg, resume treatment at 10 μg |
| | after the one-step dose increase criterion is met] |
| $\geq$ 12.0 and $\leq$ 13.0 | One-step dose reduction |
| $\geq$ 10.0 and <12.0 | Continue treatment at the current dose level* |
| ≥7.5 and <10.0 | One-step dose increase** |
| <7.5 | Discontinue treatment permanently*** and initiate another appropriate treatment |

<sup>\*</sup> If an increase of 1 g/dL is observed in 2 weeks, the dose will be reduced to the one-step lower dose level.

#### 6.5. Blinding

This will be an active-controlled, double-blind study. The study medication will be blinded through the study period to the subjects, investigator (or subinvestigator), study site staff and GSK study team. Neither the investigator (or subinvestigator) nor the subject will know which study medication the subject is receiving as all instructions regarding container number assignment and dose adjustment are given by IWRS.

#### **Roles of Person Responsible for Allocation**

The person responsible for allocation will prepare a procedure specifying the method of allocation of study treatment (study drug and control drug) and perform its duties in accordance with this document. The person responsible for allocation will confirm the indistinguishability of study treatment (study drug and control drug) and its package, and indicate the drug number on a study treatment (study drug and control drug) container. The indistinguishability of study treatment (study drug and control drug)

<sup>\*\*</sup> If an increase of >1 g/dL is observed in 2 weeks, treatment will be continued at the curent dose level. If there is a safety concern, however, the dose may be reduced at the investigator's (or subinvestigator's) discretion to the one-step lower dose level.

<sup>\*\*\*</sup> If an initial Hgb value is less than 7.5 g/dL, measurement will be repeated at the same study visit (using the same sample) to calculate the average. If the average meets the Hgb stopping criteria, study treatment will be permanently discontinued.

and its package should be checked again after completion of the study. Furthermore, the person responsible for allocation will prepare a procedure for case of an emergency that knowledge of the study treatment is essential, and break the key code of only the treatment concerned, as per request.

## **Emergency Unblinding**

- The investigator or treating physician may unblind a subject's treatment assignment only in the case of an emergency OR in the event of a serious medical condition when knowledge of the study treatment (daprodustat or darbepoetin alfa) is essential for the appropriate clinical management or welfare of the subject as judged.
- Investigators (or subinvestigators) have direct access to the subject's individual study treatment.
- It is preferred (but not required) that the investigator (or subinvestigator) first contacts the Medical Monitor or appropriate GSK study personnel to discuss options before unblinding the subject's treatment assignment.
- If GSK personnel are not contacted before the unblinding, the investigator (or subinvestigator) must notify GSK as soon as possible after unblinding, but without revealing the treatment assignment of the unblinded subject, unless that information is important for the safety of subjects currently in the study.
- The date and reason for the unblinding must be fully documented in an appropriate page of the CRF by the investigator (or subinvestigator).
- Further details of unblinding is provided in the SRM.

A subject will be withdrawn if the subject's treatment code is unblinded by the investigator (or subinvestigator). The primary reason for discontinuation (the event or condition which led to the unblinding) will be recorded in the CRF.

GSK's Global Clinical Safety and Pharmacovigilance (GCSP) staff may unblind the treatment
assignment for any subject with an SAE. If the SAE requires that an expedited regulatory report
be sent to one or more regulatory agencies, a copy of the report, identifying the subject's
treatment assignment, may be sent to investigators in accordance with local regulations and/or
GSK policy.

## 6.6. Packaging and Labeling

The contents of the label will be in accordance with all applicable regulatory requirements.

## 6.7. Preparation/Handling/Storage/Accountability

- No special preparation of study treatment is required.
- Only subjects enrolled in the study may receive study treatment and only authorized site staff
  may supply or administer study treatment. All study medications must be stored in a secure
  environmentally controlled and monitored (manual or automated) area in accordance with the
  labeled storage conditions with access limited to the investigator (or subinvestigator) and
  authorized site staff.

- Subjects must bring all of supplied study medication bottles of daprodustat/placebo at every 4 week's study visit. Study staff will collect all of study medication bottles supplied at the previous study visit and supply new study medication bottles.
- The investigator (or subinvestigator), institution, or the head of the medical institution (where applicable) is responsible for study treatment accountability, reconciliation, and record maintenance (i.e. receipt, reconciliation and final disposition records).
- Under normal conditions of handling and administration, study medication is not expected to pose significant safety risks to site staff.
- GSK will provide a document describing occupational hazards and recommended handling
  precautions either to the investigator (or subinvestigator) when necessary or upon request of the
  medical institution.
- Further details are provided in the SRM.

# 6.8. Compliance with Study Treatment Administration Daprodustat

Since daprodustat is self-administered, compliance with daprodustat treatment will be assessed through an interview with subjects at each study visit and recorded in the source document and eCRF. A record of the number of daprodustat tablets dispensed to and taken by each subject will be maintained and reconciled with study treatment and compliance records. In addition, the number of daprodustat doses dispensed, used, and unused, as well as study treatment start and stop dates will be recorded in the source document and eCRF (the number of doses returned and unreturned will also be recorded separately).

#### Darbepoetin alfa

Darbepoetin alfa will be administered to subjects once weekly at the site. Dosing details will be recorded in the source document and eCRF. Administration of darbepoetin alfa will be performed at the scheduled visit dates in principle.

## 6.9. Treatment of Study Treatment Overdose

For the purposes of this study, an overdose of daprodustat is defined as any dose greater than the highest daily dose included in the protocol. There is no specific antidote for overdose with daprodustat. The expected manifestations of daprodustat overdosage include signs and symptoms associated with an excessive and/or rapid increase in Hgb concentration. Daprodustat is highly protein bound; thus, clearance of unchanged daprodustat by hemodialysis or peritoneal dialysis is very low and these are not effective methods to enhance the elimination of daprodustat. Daprodustat metabolites are, in part, cleared via hemodialysis. In the event of a suspected overdose, it is recommended that the appropriate supportive clinical care be instituted, as dictated by the subject's clinical status. Additionally, subjects should be monitored closely for cardiovascular events, increased heart rate and hematologic abnormalities.

Consult the respective approved Prescribing Information for information on overdose for darbepoetin alfa.

## 6.10. Treatment after the End of the Study

Since the target disease studied is not life-threatening or severely debilitating and there is the alternative therapy, subjects will not receive any additional treatment from GSK after completion of the study. The investigator (or subinvestigator) is responsible for ensuring that consideration has been given to post-study care of the subject's medical condition, whether or not GSK is providing specific post-study treatment.

## 6.11. Concomitant Medications and Non-Drug Therapies

Concomitant medications, including over-the-counter medications and supplements, taken during the study will be recorded in the eCRF. Drug names and start/stop dates will be recorded for general concomitant medications, while additional details, including dose, route of administration, and dosing frequency, will be recorded for certain medications (e.g., ESAs, iron, anti-hypertensive medications). Further details are provided in the SRM.

## 6.11.1. Permitted Medications and Non-Drug Therapies

Unless specified as a prohibited medication in Section 6.11.2, all concomitant medications should be considered permitted provided they are not contraindicated for the individual subject concerned. Regular multivitamins (at recommended daily allowance) and other supplements such as calcium and vitamin D may be used if permitted by the investigator or his/her designee.

CYP2C8 is involved in the primary route of metabolism of daprodustat. Accordingly, co-administration of daprodustat with moderate CYP2C8 inhibitors (e.g., clopidogrel, teriflunomide, deferasirox) should be performed with caution.

Antihyperphosphatemic agents containing iron (e.g., ferric citrate hydrate) may be started from Week 4 onwards unless any other antihyperphosphatemic agents are appropriate. Once started, iron-containing antihyperphosphatemic agents must be continued until the end of the study wherever possible.

## 6.11.2. Prohibited Medications and Non-Drug Therapies

Use of any of the following drugs from screening until 7 days after the last dose of study treatment is prohibited:

- Strong inhibitors of CYP2C8 (e.g., gemfibrozil)
- Strong inducers of CYP2C8 (e.g., rifampin/rifampicin)

Use of the following drug; during the treatment period:

• Erythropoietin (e.g., epoetin/ darbepoetin alfa/ epoetin beta pegol)

Note: excluding darbepoetin alfa (brand name: Nesp) supplied by GSK.

## 6.12. Supplemental Iron Therapy

From Week 4, Supplemental iron therapy will be administered according to the Guidelines for Renal Anemia [The Japanese Society for Dialysis Therapy, 2016] if ferritin is  $\leq 100$  ng/mL and TSAT is  $\leq 20\%$ . The investigator (or subinvestigator) can choose the route of administration and dose of

prescription iron, and they should consider to discontinue their patient's iron therapy if ferritin is ≥300 ng/mL [The Japanese Society for Dialysis Therapy , 2016]. Refer to 4.2. regading iron use until Week 4.

## 7. Study Assessments and Procedures

Protocol waivers or exemptions are not allowed with the exception of immediate safety concerns. Therefore, adherence to the study design requirements, including those specified in the Time and Events Table, are essential and required for study conduct.

## 7.1. Time and Events Table

The time and events tables for the entire study and PK assessment are presented as Table 10 and Table 11, respectively. Throughout the study period, including the screening, treatment and follow-up periods, the study visit days should occur on the first dialysis session day of the week (e.g., if Monday-Wednesday-Friday schedule, the study visit should be on Monday) and Visit days will be counted from Day 1. To allow for a flexible schedule, the allowable window for Screening Visit will be "2-4 weeks  $\pm$  3 days prior to Day 1", and that for the visits after Day 1 will be " $\pm$  3 days". In any case, the study visit should occur on the first dialysis session day of the week. Unless otherwise specified, all assessments should occur before dialysis on the day.

Table 10 Time and Events Table

| Phase | Screening | Treatment | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | -4~-2 <sup>11</sup> | Day 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20 | 22 | 24 | 26 | 28 |
| All assessments pre-dialysis, unless noted. Allowance range (days) | ±3 | _ | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 |
| | | - | 3 | 3 | <u> </u> | -3 | -3 | | 3 | 3 | -3 | -3 | <u> </u> | -3 | | 3 |
| Informed consent | X | | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria | X | X | | | | | | | | | | | | | | |
| Medical history, demography, height <sup>1</sup> , weight <sup>1</sup> | X | | | | | | | | | | | | | | | |
| Registration with IWRS | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Study medication dispensing <sup>2, 3</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Study treatment compliance | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Vital signs (before and after dialysis) 4 | X | X | | X | | | | | | X | | | | | | X |
| Ophthalmology <sup>5</sup> | X <sup>12</sup> | | | | | | • | | <b>—</b> | | | | | | | |
| ECG | X | | | | | | | | | | | | | X | | |
| HemoCue Hgb | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Hematology | X | X | | X | | Hgb<br>only | | Hgb<br>only | | X | | Hgb<br>only | | Hgb<br>only | | X |
| Clinical chemistry | X | X | | X | | | | | | X | | | | | | X |
| Pregnancy test (serum hCG) <sup>6</sup> | X | X | | X | | | | | | X | | | | | | X |
| Estradiol, FSH <sup>7</sup> | X | | | | | | | | | | | | | | | |
| PK <sup>8</sup> | | | | | | | | X | | | | | | X | | |
| Ferritin, TSAT | X | X | | X | | | | | | X | | | | | | X |
| Serum iron, TIBC, UIBC, serum transferrin, hepcidin | | X | | X | | | | | | X | | | | | | X |
| iPTH | | X | | | | | | | | | | | | | | X |
| HR-QoL (SF-36, EQ-5D-5L/ EQ-VAS) | | X | | | | | | X | | | | | | | | X |
| Genetics sample 9 | | X | | | | | | | | | | | | | | |
| AE assessment 10 | X 13 | - | | | | | | | | | | | | | | <b>→</b> |
| Concomitant Medications Review | - | | | | | | | | | | | | | | | <b>→</b> |
| Phase | | | | | | | Treatmo | ent | | | | | | Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit All assessments pre-dialysis, unless noted. | 30 | 32 | 34 | 36 | 38 | 40 | 42 | 44 | 46 | 48 | 50 | 52 | Early<br>withdrawal | 2 weeks<br>after Week 52<br>or early<br>withdrawal |
| Allowance range (days) | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | ±3 | - | ±3 |
| Informed consent | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria | | | | | | | | | | | | | | |
| Medical history, demography, height <sup>1</sup> , weight <sup>1</sup> | | | | | | | | | | | | | | |
| Registration with IWRS | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Study medication dispensing <sup>2, 3</sup> | X | X | X | X | X | X | X | X | X | X | X | | | |
| Study treatment compliance | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Vital signs (before and after dialysis) 4 | | | | | | X | | | | | | X | X | X |
| Ophthalmology <sup>5</sup> | | | | | | | | | | - | | <b></b> | $\leftarrow$ | |
| ECG | | | | | | | | | | | | X | | |
| HemoCue Hgb | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Hematology | | Hgb<br>only | | Hgb<br>only | | X | | Hgb<br>only | | Hgb<br>only | | X | X | X |
| Clinical chemistry | | | | | | X | | | | | | X | X | X |
| Pregnancy test (serum hCG) 6 | | | | | | X | | | | | | X | X | X |
| Estradiol, FSH <sup>7</sup> | | | | | | | | | | | | | | |
| PK 8 | | | | | | | | | | | | | | |
| Ferritin, TSAT | | | | | | X | | | | | | X | X | |
| Serum iron, TIBC, UIBC, serum transferrin, hepcidin | | | | | | X | | | | | | X | X | |
| iPTH | | | | | | | | | | | | X | | |
| HR-QoL | | | | | | | | | | | | X | X | |
| Genetics sample 9 | | | | | | | | | | | | | | |
| AE assessment 10 | <del></del> | | | | | | | | | | | | | <b>—</b> |
| Concomitant Medications Review | <b>←</b> | | | | | | | | | | | | | <u> </u> |

<sup>1.</sup> Body weight is measured after dialysis. Both height and body weight are measured only at screening.

<sup>2.</sup> Daprodustat/placebo will be dispensed once every 4 weeks, and darbepoetin alfa/placebo will be dispensed once every 2 weeks

<sup>3.</sup> If a subject visit the study site only to receive study medication, only registration with the IWRS study medication dispensing, and study medication compliance will be required.

2015N266251\_02 **CONFIDENTIAL** PHI201754

- 4. At visits without dialysis, only one measurement of each parameter will be obtained.
- 5. Ophthalmology exams should be conducted at the following time points.
  - Screening: anytime after consenting and prior to first dose of study medication (Day 1)
  - Week 12: window from weeks 10-14 (inclusive)
  - End of study: window from weeks 48-52 (inclusive)
  - Early study medication discontinuation: withdrawal eye exam as close to the last dose as possible (the repeat exams are not required if one has been performed within the 2 prior weeks).
- 6. Performed in females of childbearing potential.
- 7. Measured in female subjects only to determine the menopausal status (see Section 5.1.)
- 8. See Table 11.
- 9. Informed consent for optional Genetic research should be obtained before collecting a sample (see Section 7.6.).
- 10. See Section7.4.1.1..
- 11. The interval between screening and Day 1 should be 4 weeks in subjects treated with epoetin beta pegol every 4 weeks or darbepoetin alfa every 4 weeks in the prior ESA therapy.
- 12. For re-screening subjects, no repeated ophthalmology exams could be required at re-screening, in which case the results of ophthalmology exams at the most recent screening could be replaced on the investigator's (or subinvestigator's) discretion if re-screening subjects meet all of the following criteria:
  - There were no findings that would suggest a repeat ophthalmology exam performed within the next 3 months at the latest screening ophthalmology exam.
  - No new ocular symptoms or complaints were noted after the most recent ophthalmologic screening and before the next re-screening.
  - The most recent ophthalmology screening was performed within 3 months prior to anticipated Day 1.
- 13. Only SAEs assessed as related to study participation or a GSK product are collected.
- 14. For withdrawn subjects, specified assessments should be done wherever possible.

Table 11 Blood Sampling Schedule for Pharmacokinetics

| PK sample | Week 12 <sup>2</sup> | Week 24 <sup>2</sup> |
|---|---|---|
| Blood sampling timing <sup>1</sup> | 1, 2, 3, and 4 h after administration of daprodustat or placebo | |

Subjects must take the study medication with regard to blood sampling time. Subjects will record the date and time of the last two study medication doses taken prior to blood sampling in the medication diary. There should be an interval of at least 12h (preferably, almost 24 h) between these two doses.

- 1. Blood sampling should be completed within +/- 30 min of the planned collected time.
- 2. Blood sampling not performed at this visit may be postponed until the following visits.

#### 7.2. Screening and Critical Baseline Assessments

Cardiovascular medical history/risk factors will be assessed (documented in the eCRF) at baseline. In addition, the following demographic information will be collected:

- Year of birth
- Gender
- Race and ethnic
- Medical history/treatment history/family history will be assessed in relation to the inclusion/exclusion criteria (Section 5.1, 5.2).

Full details of baseline assessments are provided in Time and Events Table (Table 10).

## 7.3. Efficacy

Efficacy will be assessed according to the Time and Event Table (Table 10).

Hgb concentrations measured by the central laboratory will be mainly used for efficacy assessment. GSK will supply a point-of-care Hgb analyzer (HemoCue) to each site for rapid and convenient measurement of Hgb and to ensure consistency of Hgb measurements across all sites participating in the study. Assessment for Hgb concentrations via HemoCue will be used for eligibility (Section 5.1), permanent discontinuation of study treatment (Section 5.4), and dose adjustment criteria (Section 6.4). In addition, assessments of iron metabolism parameters used for exploratory assessment is outlined with specific procedures in Section 7.4.7.

#### 7.4. Safety

Planned time points for all safety assessments are listed in the Time and Events Table (Table 10). Additional time points for safety tests (such as vital signs, physical exams and laboratory safety tests) may be added during the course of the study based on newly available data to ensure appropriate safety monitoring

#### 7.4.1. Adverse Events (AE) and Serious Adverse Events (SAEs)

The definitions of an AE or SAE can be found in Section 12.6. Appendix 6.

The investigator and their designees are responsible for detecting, documenting and reporting events that meet the definition of an AE or SAE.

# 7.4.1.1. Time period and Frequency for collecting AE and SAE information

• AEs and SAEs will be collected from the start of Study Treatment until the follow-up contact (see Section 7.4.1.3.), at the timepoints specified in the Time and Events Table (Table 10).

- Medical occurrences that begin prior to the start of study treatment but after obtaining informed consent may be recorded on the Medical History/Current Medical Conditions section of the CRF.
- Any SAEs assessed as related to study participation (e.g., protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK product will be recorded from the time a subject consents to participate in the study up to and including any follow-up contact.
- All SAEs will be recorded and reported to GSK within 24 hours, as indicated in Section 12.6.
   Appendix 6.
- Investigators are not obligated to actively seek AEs or SAEs in former study subjects. However, if the investigator learns of any SAE, including a death, at any time after a subject has been discharged from the study, and he/she considers the event reasonably related to the study treatment or study participation, the investigator must promptly notify GSK.

NOTE: The method of recording, evaluating and assessing causality of AEs and SAEs plus procedures for completing and transmitting SAE reports to GSK are provided in Section 12.6. Appendix 6.

#### 7.4.1.2. Method of Detecting AEs and SAEs

Care will be taken not to introduce bias when detecting AEs and/or SAEs. Open-ended and non-leading verbal questioning of the subject is the preferred method to inquire about AE occurrence. Appropriate questions include:

- "How are you feeling?"
- "Have you had any (other) medical problems since your last visit/contact?"
- "Have you taken any new medicines, other than those provided in this study, since your last visit/contact?"

#### 7.4.1.3. Follow-up of AEs and SAEs

After the initial AE/SAE report, the investigator is required to proactively follow each subject at subsequent visits/contacts. All SAEs, and non-serious AEs of special interest (as defined in Section 7.4.2.) will be followed until resolution, until the condition stabilizes, until the event is otherwise explained, or until the subject is lost to follow-up (as defined in Section 5.4.). Further information on follow-up procedures is given in Section 12.6. Appendix 6...

#### 7.4.1.4. Cardiovascular and Death Events

For any cardiovascular events detailed in Section 12.6. Appendix 6 and all deaths, whether or not they are considered SAEs, specific Cardiovascular (CV) and Death sections of the CRF will be required to be completed. These sections include questions regarding cardiovascular (including sudden cardiac death) and non-cardiovascular death.

The CV CRFs are presented as queries in response to reporting of certain CV Medical Dictionary for Regulatory Activities (MedDRA) terms. The CV information should be recorded in the specific cardiovascular section of the CRF within one week of receipt of a CV Event data query prompting its completion.

The Death CRF is provided immediately after the occurrence or outcome of death is reported. Initial and follow-up reports regarding death must be completed within one week of when the death is reported.

#### 7.4.1.5. Regulatory Reporting Requirements for SAEs

Prompt notification by the investigator to GSK of SAEs and non-serious AEs related to study treatment (even for non- interventional post-marketing studies) is essential so that legal obligations and ethical responsibilities towards the safety of subjects and the safety of a product under clinical investigation are met.

GSK has a legal responsibility to notify both the local regulatory authority and other regulatory agencies about the safety of a product under clinical investigation. GSK will comply with country specific regulatory requirements relating to safety reporting to the regulatory authority, Institutional Review Board (IRB)/Independent Ethics Committee (IEC) and investigators.

Investigator safety reports are prepared for suspected unexpected serious adverse reactions according to local regulatory requirements and GSK policy and are forwarded to investigators as necessary.

An investigator who receives an investigator safety report describing a SAE(s) or other specific safety information (e.g., summary or listing of SAEs) from GSK will file it with the IB and will notify the IRB/IEC, if appropriate according to local requirements.

## 7.4.2. Adverse Events of Special Interest

The investigator (or subinvestigator) or designee will be responsible for detecting, documenting, and reporting any AEs of special interest listed below. These events have been identified based on the known safety profiles of ESAs, theoretical or potential risks based on the mechanism of action of daprodustat, and findings from completed nonclinical studies of daprodustat.

- Thrombosis and/or tissue ischemia secondary to excessive erythropoiesis
- Death, myocardial infarction, stroke, heart failure, thromboembolic events, thrombosis of vascular access
- Cardiomyopathy
- Pulmonary artery hypertension (PAH)
- Cancer-related mortality and tumor progression and recurrence
- Esophageal and gastric erosions
- Proliferative retinopathy, macular edema, choroidal neovascularization
- Exacerbation of rheumatoid arthritis

Any relevant AE should be recorded in the relevant section of the subject's eCRF.

#### 7.4.3. Pregnancy

• Details of all pregnancies in female subjects will be collected after the start of dosing and until the follow-up contact.

• If a pregnancy is reported then the investigator should inform GSK within 2 weeks of learning of the pregnancy and should follow the procedures outlined in Section 12.4. Appendix 4.

#### 7.4.4. Medical Device Incidents (Including Malfunctions)

The medical devices (i.e., the darbepoetin alfa plastic prefilled syringes) are being provided for use in this study. The investigator is responsible for the detection and documentation of events meeting the definitions of incident or malfunction that occur during the study with such devices.

The definition of a Medical Device Incident can be found in Appendix 8 (Section 12.8.)

NOTE: Incidents fulfilling the definition of an AE/SAE will also follow the processes outlined in Section 7.4.1. and Appendix 6 (Section 12.6) of the Protocol.

#### 7.4.4.1. Time Period for Detecting Medical Device Incidents

- Medical device incidents or malfunctions of the device that result in an incident will be detected, documented and reported during all periods of the study in which the medical devices are available for use.
- If the investigator learns of any incident at any time after a subject has been discharged from the study, and such incident is reasonably related to a medical device provided for the study, the investigator will promptly notify GSK. NOTE: The method of documenting Medical Device Incidents is provided in Appendix 8 (Section 12.8).

# 7.4.4.2. Follow-up of Medical Device Incidents

- All medical device incidents involving an AE, will be followed until resolution of the event, until the condition stabilizes, until the condition is otherwise explained, or until the subject is lost to follow-up (as defined in Section 5.4.). This applies to all subjects, including those withdrawn prematurely.
- The investigator is responsible for ensuring that follow-up includes any supplemental
  investigations as may be indicated to elucidate as completely as practical the nature and/or
  causality of the incident.
- New or updated information will be recorded on the originally completed form "Medical Device Incident Report Form" with all changes signed and dated by the investigator.

#### 7.4.4.3. Prompt Reporting of Medical Device Incidents to GSK

- Medical device incidents will be reported to GSK within 24 hours once the investigator determines that the event meets the protocol definition of a medical device incident.
- Facsimile transmission of the "Medical Device Incident Report Form" is the preferred method to transmit this information to the SAE contact information.
- The same individual will be the contact for receipt of medical device reports and SAEs.
- In the absence of facsimile equipment, notification by telephone is acceptable for incidents, with a copy of the "Medical Device Incident Report Form" sent by overnight mail.

#### 7.4.5. Vital Signs/Height/Weight

Systolic and diastolic blood pressure and heart rate will be measured before and after dialysis, in sitting or semi-supine position (chair for dialysis is acceptable) after at least 5 minutes rest. When measuring before dialysis, it should be conducted prior to blood sampling for lab tests. One reading of blood pressure and heart rate will be taken and recorded in the source document and the CRF. Height and weight will be measured at screening visit only. Weight should be measured after dialysis.

# 7.4.6. Electrocardiogram (ECG)

12-lead ECGs will be recorded in supine position. The heart rate, PR, QRS, and QT (pre-corrected) intervals will be measured. QTcB should be calculated by machine or manually by designated staff at each site. The investigator determines whether the ECG data is assessable or not. Measurement method and measurement timing (i.e., before or after dialysis) should be consistent as far as possible during the study period.

At Screening visit when an ECG is performed, two additional ECGs are required if initial ECG indicates prolonged QTc. The average QTcB value of all three ECGs will be used to determine eligibility.

QTc exclusion criteria can be found in Section 5.2. Refer to SRM for further details.

# 7.4.7. Clinical Laboratory Assessments

All study-required laboratory assessments will be performed by a central laboratory with the exception of HemoCue Hgb. The results of each HemoCue Hgb must be entered into the subject's eCRF. Details are provided in the SRM.

All laboratory assessments, as defined in Table 12, must be conducted in accordance with the Laboratory Manual and Protocol Time and Events Schedule (Table 10). Laboratory requisition forms must be completed and samples must be clearly labeled with the subject number, protocol number, site/center number, and sample collection date. Reference ranges for all parameters will be provided to the site by the central laboratory. Details of blood sampling (including the volume of blood to be collected) as well as procedures for processing, storage, and shipment of samples are provided in the SRM.

PK assessment of daprodustat is outlined in Section 7.5.

| Laboratory assessment | | Parameter | |
|---|---|---|---|
| | Platelet count | RBC indices: | WBC dfferential |
| | RBC count | MCV | Neutrophils |
| Hamatalagu | Reticulocyte count | MCH | Lymphocytes |
| Hematology | Hemoglobin | MCHC | Monocytes |
| | Hematocrit | RDW | Eosinophils |
| | WBC count | | Basophils |
| | Sodium | AST | Bicarbonate |
| | Potassium | ALT | Inorganic phosphate |
| | Chloride | Creatinine | Glucose |
| Clinical chemistry | Calcium (total and albumin-<br>corrected) | Total bilirubin | Direct/indirect bilirubin |
| | Albumin | Urea nitrogen | |
| | Total cholesterol | HDL cholesterol | LDL cholesterol |
| | Serum iron | Serum ferritin | Serum transferrin |
| Iron parameters | TIBC | UIBC | TSAT |
| | Hepcidin | | |
| Other laboratory | FSH <sup>1</sup> | Estradiol 1 | iPTH |
| tests | serum hCG <sup>2</sup> | | |

Table 12 Laboratory Assessments

If additional non-protocol specified laboratory assessments are performed at the institution's local laboratory and result in a change in subject management or are considered clinically significant by the investigator (or subinvestigator) (e.g., SAE or AE or dose modification), the results must be recorded in the eCRF.

Refer to the SRM for appropriate processing and handling of samples to avoid duplicate and/or additional blood draws.

All laboratory tests with values that are considered clinically significantly abnormal during participation in the study should be repeated until the values return to normal or baseline. If such values do not return to normal within a period judged reasonable by the investigator (or subinvestigator), the etiology should be identified and the Sponsor notified.

#### 7.4.8. Ophthalmology

Ophthalmology exams will be performed by a study-designated ophthalmology specialist. Each assessment will include a comprehensive eye exam with at least the following components: measurement of best corrected visual acuity, intraocular pressure, an anterior chamber exam, and a fundoscopic exam. These exams will be used for assessment of ocular adverse events. Assessment results will be captured on worksheets which will be transferred to the eCRF. Additional details on the process for completing these assessments are provided in the SRM.

#### 7.5. Pharmacokinetics

Blood samples for PK analysis of daprodustat will be collected as outlined in Table 11, and the date and time of the last two study medication doses taken prior to blood sampling as well as the date and time of sampling must be recorded in the eCRF.

<sup>1.</sup> Measured in female subjects only to determine the menopausal status (see Section 5.1).

<sup>2.</sup> Performed in females of childbearing potential.

Blood PK analysis will be performed under the control of GSK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics (PTS-DMPK)/Scinovo and GSK-Japan Bioanalysis, the details of which will be included in the SRM. Concentrations of parent daprodustat will be determined in blood samples using the currently established analytical methodology. Raw data will be archived at the bioanalytical site.

Procedures for processing, storage, and shipment of samples are provided in the SRM.

#### 7.6. Genetics

A blood sample will be collected for genetic analysis from consenting subjects. This sample can be collected on Day 1 once written informed consent has been obtained. Information regarding genetic research is included in Section 12.7. Appendix 7.

# 7.7. Patient Reported Outcome (PRO)

The patient reported outcome (PRO) [e.g.health-related QOL (HRQoL), health status and health utility] will be assessed using several rating scales.

All questionnaires used in this study have been translated into Japanese and are validated and will be administered in paper version.

Specific instructions on how the subject is to complete the scales and the process for data entry are provided in the SPM.

#### 7.7.1. Health Related Quality of Life (SF-36)

The SF-36 acute version is a general health status questionnaire designed to elucidate the patient's perception of his/her health on several domains, including physical functioning, role physical, bodily pain, vitality, social functioning, role emotional, mental health, and general health over the past seven days. The questionnaire contains 36 Likert type questions that ask the patient to recall how he/she felt during the past seven days.

•

# 7.7.2. EuroQol 5 Dimension 5 Level Health Utility Index (EQ-5D-5L)/ EuroQol Visual Analogue Scale (EQ-VAS)

The EQ-5D-5L is intended to measure the general health status and health utility. The EQ-5D-5L consists of 2 concepts: self-reported health status consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses (no problems/slight problems/moderate problems/severe problems/extreme problems) and self-rated health utility on a visual analogue scale (VAS), from 'best imaginable health state' and 'worst imaginable health state'.

#### 8. DATA MANAGEMENT

- For this study subject data will be entered into GSK defined CRFs, transmitted electronically to GSK or designee and combined with data provided from other sources in a validated data system.
- Management of clinical data will be performed in accordance with applicable GSK standards and data cleaning procedures to ensure the integrity of the data, e.g., removing errors and inconsistencies in the data.
- Adverse events and concomitant medications terms will be coded using MedDRA and an internal validated medication dictionary, GSKDrug.
- CRFs (including queries and audit trails) will be retained by GSK, and copies will be sent to the
  investigator to maintain as the investigator copy. Subject initials will not be collected or
  transmitted to GSK according to GSK policy.

#### 9. STATISTICAL CONSIDERATIONS AND DATA ANALYSES

A detailed description of any planned analyses will be documented in a RAP. Any deviations from the analyses described in the protocol will be documented in the RAP or the final study report.

#### 9.1. Hypotheses

The primary objective of the study is to demonstrate the non-inferiority of daprodustat to darbepoetin alfa based on mean Hgb during the primary efficacy evaluation period (Weeks 40 to 52) in HD subjects. As a preliminary assessment, it will be confirmed whether the lower and upper limit of 95% CI for mean Hgb during the primary efficacy evaluation period in daprodustat group would be in target range (10.0-12.0 g/dL) at first. And then the following non-inferiority statistical hypotheses are to be tested at a one-sided significance level of 2.5% (i.e. two-sided significance level of 5%):

- H<sub>0</sub>: Treatment difference in mean Hgb during the primary efficacy evaluation period is -1.0 g/dL or less
- H<sub>1</sub>: Treatment difference in mean Hgb during the primary efficacy evaluation period is greater than -1.0 g/dL.

Only when the primary endpoint achieves non-inferiority, statistical testing will progress to the principal secondary endpoint with a focus on superiority according to the step-down procedure. More specifically, the superiority of daprodustat to darbepoetin alfa in terms of target Hgb control in HD subjects is to be demonstrated at a two-sided significance level of 5% by testing the following statistical hypotheses:

- H<sub>0</sub>: The proportion of subjects whose mean Hgb during the primary efficacy evaluation period is within the target range (10.0-12.0 g/dL) is equal between the treatment groups.
- H<sub>1</sub>: The proportion of subjects whose mean Hgb during the primary efficacy evaluation period is within the target range (10.0-12.0 g/dL) is different between the treatment groups.

#### 9.2. Sample Size Considerations

#### 9.2.1. Sample Size Assumptions

Assuming a non-inferiority margin of -1.0 g/dL, a treatment difference of 0.0 g/dL, and a standard deviation of 1.5 g/dL for mean Hgb during the primary efficacy evaluation period in HD subjects, two-sample t-test has at least 99% power at a one-sided significance level of 2.5% (i.e. two-sided significance level of 5%) with a sample size of 100 subjects per group. Assuming a dropout rate of approximately 25%, 135 subjects will be randomized to each group. Given the results from previous non-inferiority studies of similar drugs (darbepoetin alfa, epoetin beta pegol, and peginesatide), the non-inferiority margin of -1.0 g/dL is set. Since an increase of 1.0 g/dL indicates improvement in anemia according to the guidelines for renal anemia in Japan, the non-inferiority margin of -1.0 g/dL may be the clinically acceptable largest difference in renal anemia.

While the present study is designed to ensure long-term safety data from 100 HD subjects, and the primary hypothesis test has at least 99% power to estimate the efficacy very precisely, non-inferiority can be statistically demonstrated with a minimum between-group difference of -0.582 g/dL.

# 9.2.2. Sample Size Sensitivity

The power is shown according to treatment difference and standard deviation in Table 13.

Table 13 Power Sensitivity (100 Subjects Evaluated, Noninferiority Margin of -1.0, One-Sided Significance Level of 2.5%)

| Treatment | | Standard deviation | |
|------------|--------|--------------------|-------|
| difference | 1.25 | 1.5 | 1.75 |
| 0 | 100.0% | 99.7% | 98.0% |
| -0.1 | 99.9% | 98.8% | 95.1% |
| -0.2 | 99.5% | 96.4% | 89.6% |
| -0.3 | 97.6% | 90.7% | 80.4% |

#### 9.2.3. Sample Size Re-estimation or Adjustment

No sample size re-estimation is planned for this study.

#### 9.3. Data Analysis Considerations

#### 9.3.1. Analysis Populations

• All Screening Population

The All Screening Population consists of all subjects who are given subject number and whose data are collected, including demographics at screening.

#### • Intention-To-Treat (ITT) Population

The ITT Population consists of all subjects who are given a randomization number regardless of whether they actually receive study treatment and whose Hgb assessment was performed at baseline and at least one scheduled post-baseline visit. Subjects will be analyzed according to randomized treatment. This population will be the primary population for an assessment of non-inferiority.

• modified ITT (mITT) Population

The mITT Population consists of all ITT subjects who have at least one Hgb measurement during the efficacy evaluation period. Subjects will be analyzed according to randomized treatment. This population will be the primary population for an assessment of superiority.

#### • Per-Protocol (PP) Population

The PP Population consists of all mITT subjects who are not major protocol violators. Details will be defined in the RAP. This population will be used for efficacy sensitivity analyses.

#### Safety Population

The Safety Population consists of subjects who receive at least one dose of study treatment. Subjects will be analyzed according to the treatment received. This population will be used for safety analyses.

#### • PK Population

The PK Population consists of all daprodustat -treated subjects from whom PK samples are collected and analyzed.

Additional populations may be defined in the RAP.

#### 9.3.2. Interim Analysis

No interim analysis is planned.

#### 9.3.3. Adjustment for Multiplicity

Adjustment for multiplicity will be applied to maintain an overall type I error rate of 5%. After a preliminary assessment, the primary endpoint will be evaluated to demonstrate the non-inferiority at a one-sided significance level of 2.5% (i.e. two-sided significance level of 5%). Only when the primary endpoint achieves non-inferiority, statistical testing will progress to the principal secondary endpoint with a focus on superiority. Since the process will follow step-down manner, a multiplicity adjustment will not be needed according to a closed test procedure, similarly two-sided significance level of 5% will be used.

Other secondary endpoints, which will be evaluated on a complementary or exploratory basis, will be compared at a two-sided significance level of 5% without multiplicity adjustment.

#### 9.4. Key Elements of Analysis Plan

#### 9.4.1. Primary Efficacy Analysis

The primary endpoint, which is the mean Hgb during the primary efficacy evaluation period, will be analyzed to demonstrate the non-inferiority of daprodustat to darbepoetin alfa in HD subjects. MMRM will be used to estimate the mean Hgb during the primary efficacy evaluation period and its 95% CI by treatment groups. This model includes treatment groups, baseline Hgb, assessment visits, interaction terms between treatment groups and assessment visits, as well as interaction terms between baseline Hgb and assessment visit. As a preliminary assessment, it will be confirmed if the lower and upper limit of 95% CI for mean Hgb during the primary efficacy evaluation period in daprodustat group would be in target range (10.0- 12.0 g/dL) at first. This confirmation will be established if the lower and upper limit of 95% CI for the mean Hgb in daprodustat group based on observed Hgb

would lie fully within target range (10.0-12.0 g/dL). In addition, the point estimate and 95% CI for the treatment difference (daprodustat - darbepoetin alfa) in the mean Hgb during the primary efficacy evaluation period will be estimated. Non-inferiority will be established if the lower limit of the 95% CI is greater than -1.0 g/dL. Even if the 95% CI for the difference is completely negative (i.e. lies fully within the range -1.0 to <0 g/dL) non-inferiority would still be concluded on condition that the mean Hgb estimated in the daprodustat group is within the target range.

The primary efficacy population will be the ITT Population, and the analysis will be repeated in the mITT and PP Population to evaluate the robustness of the conclusion. Following sensitivity analyses will be conducted to assess robustness of study result.

- If there are Hgb considered to be impacted by blood transfusion or marketed rhEPO/ESAs, sensitivity analysis excluding the Hgb values from the analyses of primary endpoint will be conducted.
- Analysis of covariance (ANCOVA) will be conducted as sensitivity analysis to MMRM. This
  model includes treatment group and baseline Hgb. The analysis population will be mITT
  population and the similar analysis will be repeated in the PP population.
- A tipping point analysis based on multiple imputation will be conducted as sensitivity analysis to
  missing data assumption. This analysis explores a point where non-inferiority is not confirmed
  (tipping point) by changing assumption to missing data and repeating imputation. The analysis
  population will be ITT population and the similar analysis will be repeated in the mITT and PP
  population.

Further details of sensitivity analyses will be provided in the RAP.

# 9.4.2. Principal Secondary Efficacy Analysis

The principal secondary endpoint, which is the proportion of subjects whose mean Hgb during the primary efficacy evaluation period is within the target range, will be analyzed to demonstrate the superiority of daprodustat to darbepoetin alfa in HD subjects.

In the mITT Population, a logistic regression model including treatment group and baseline Hgb as covariates will be used to estimate the point estimate and 95% CI for the odds ratio (daprodustat/darbepoetin alfa). This analysis will be performed to demonstrate the superiority at a two-sided significance level of 5%, conditional on the primary endpoint achieving noninferiority. Superiority will be established if the lower limit of the 95% CI for odds ratio is greater than 1.0.

#### 9.4.3. Other Secondary Efficacy Analyses

Among the secondary efficacy endpoints, the time (%) in Hgb target range during the primary efficacy evaluation period , and proportion of subjects who have an Hgb increase of more than 2 g/dL over any 4 weeks, the point estimates and 95% CIs for the treatment difference (or odds ratio) in HD subjects will be calculated. Other secondary efficacy and exploratory endpoints will be summarized by each treatment group.

#### 9.4.4. Safety Analyses

In principle, safety data will be summarized by each treatment group in the Safety Population.

#### 9.4.4.1. Exposure

Exposure information will be listed for all subjects. The duration of treatment (number of days) and cumulative dose will be tabulated. In addition, distribution of the dose level at each assessment visit and final dosing visit will be tabulated. Frequency of dose adjustment and duration of treatment interruption due to Hgb >13.0 g/dL will be summarized.

#### 9.4.4.2. Adverse Events

All AEs will be categorized by the MedDRA system organ class and preferred term to tabulate the number and incidence. All AEs, SAEs, AEs leading to discontinuation of study treatment, and AEs of special interest will be summarized separately. Similar summary will be provided for study treatment-related AEs.

#### 9.4.4.3. Other Safety Parameters

For laboratory tests, vital signs and ECG, parameters and/or changes from baseline will be summarized using summary statistics at each assessment visit. The number and percentage of subjects with values of the potential clinical importance values will be tabulated. The criteria for the potential clinical importance will be described in the RAP. For lipid parameters (total cholesterol, LDL cholesterol, and HDL cholesterol), percent changes will also be tabulated. The number (%) of subjects who have any change in anti-hypertensive medications (type and/or dose) due to increased blood pressure will be tabulated.

#### 9.4.5. Pharmacokinetics Analyses

For plasma concentrations of daprodustat over time, individual data will be listed, and summary statistics at each time point will be calculated for each dose level. For PK parameters (AUC <sub>0-4</sub> and Cmax), summary statistics will be calculated for each dose level, and scatter plots against the dose level will be generated.

#### 9.4.6. PRO Data Analysis

Details of PRO data tabulation will be described in the RAP.

#### 10. STUDY GOVERNANCE CONSIDERATIONS

#### 10.1. Posting of Information on Publicly Available Clinical Trial Registers

Study information from this protocol will be posted on publicly available clinical trial registers before enrollment of subjects begins.

# 10.2. Regulatory and Ethical Considerations, Including the Informed Consent Process

The study will be conducted in accordance with "the Ministerial Ordinance on the Standards for the Conduct of Clinical Trials of Medicinal Products (MHW Notification No.28 dated 27th March, 1997)" and the Pharmaceutical Affairs Law.

GSK will submit the CTN to the regulatory authorities in accordance with with Article 80-2 of the Pharmaceutical Affairs Law before conclusion of any contract for the conduct of the study with study sites.

The study will be conducted in accordance with all applicable regulatory requirements, and with GSK policy.

The study will also be conducted in accordance with ICH Good Clinical Practice (GCP), all applicable subject privacy requirements, and the guiding principles of the current version of the Declaration of Helsinki. This includes, but is not limited to, the following:

- IRB/IEC review and favorable opinion/approval of the study protocol and amendments as applicable
- Signed informed consent to be obtained for each subject before participation in the study (and for amendments as applicable)
- Investigator reporting requirements (e.g. reporting of AEs/SAEs/protocol deviations to IRB/IEC)
- GSK will provide full details of the above procedures, either verbally, in writing, or both.
- The IEC/IRB, and where applicable the regulatory authority, approve the clinical protocol and all optional assessments, including genetic research.
- Optional assessments (including those in a separate protocol and/or under separate informed consent) and the clinical protocol should be concurrently submitted for approval unless regulation requires separate submission.
- Approval of the optional assessments may occur after approval is granted for the clinical protocol
  where required by regulatory authorities. In this situation, written approval of the clinical
  protocol should state that approval of optional assessments is being deferred and the study, with
  the exception of the optional assessments, can be initiated.

#### **Informed Consent**

Prior to participation in the study, the investigator (or subinvestigator) should fully inform the potential subject and the subject's legally acceptable representative (as required) of the study including the written information. The investigator (or subinvestigator) should provide the subject and the subject's legally acceptable representative ample time and opportunity to inquire about details of the study. The subject and the subject's legally acceptable representative should sign and personally date the consent form. If the subject wishes to consider the content of the written information at home,

he/she may take the consent form home. The person who conducted the informed consent discussion and study collaborator giving supplementary explanation, where applicable, should sign and personally date the consent form. If an impartial witness is required, the witness should sign and personally date the consent form. The investigator (or subinvestigator) should retain this signed and dated form (and other written information) together with the source medical records, such as clinical charts (in accordance with the rules for records retention, if any, at each medical institution) and give a copy to the subject and the subject's legally acceptable representative.

## 10.3. Quality Control (Study Monitoring)

- In accordance with applicable regulations including GCP, and GSK procedures, GSK monitors will contact the site prior to the start of the study to review with the site staff the protocol, study requirements, and their responsibilities to satisfy regulatory, ethical, and GSK requirements.
- When reviewing data collection procedures, the discussion will also include identification, agreement and documentation of data items for which the CRF will serve as the source document.

GSK will monitor the study and site activity to verify that the:

- Data are authentic, accurate, and complete.
- Safety and rights of subjects are being protected.
- Study is conducted in accordance with the currently approved protocol and any other study agreements, GCP, and all applicable regulatory requirements.

•

The investigator and the head of the medical institution (where applicable) agrees to allow the monitor direct access to all relevant documents

#### 10.4. Quality Assurance

- To ensure compliance with GCP and all applicable regulatory requirements, GSK may conduct a quality assurance assessment and/or audit of the site records, and the regulatory agencies may conduct a regulatory inspection at any time during or after completion of the study.
- In the event of an assessment, audit or inspection, the investigator (and institution) must agree to grant the advisor(s), auditor(s) and inspector(s) direct access to all relevant documents and to allocate their time and the time of their staff to discuss the conduct of the study, any findings/relevant issues and to implement any corrective and/or preventative actions to address any findings/issues identified.

#### 10.5. Study and Site Closure

- Upon completion or premature discontinuation of the study, the GSK monitor will conduct site
  closure activities with the investigator or site staff, as appropriate, in accordance with applicable
  regulations including GCP, and GSK Standard Operating Procedures.
- GSK reserves the right to temporarily suspend or prematurely discontinue this study at any time for reasons including, but not limited to, safety or ethical issues or severe non-compliance. For
- multicenter studies, this can occur at one or more or at all sites.

- If GSK determines such action is needed, GSK will discuss the reasons for taking such action with the investigator or the head of the medical institution (where applicable). When feasible, GSK will provide advance notification to the investigator or the head of the medical institution, where applicable, of the impending action.
- If the study is suspended or prematurely discontinued for safety reasons, GSK will promptly inform all investigators, heads of the medical institutions (where applicable) and/or institution(s) conducting the study. GSK will also promptly inform the relevant regulatory authorities of the suspension or premature discontinuation of the study and the reason(s) for the action.
- If required by applicable regulations, the investigator or the head of the medical institution (where applicable) must inform the IRB/IEC promptly and provide the reason for the suspension or premature discontinuation.

#### 10.6. Records Retention

- Following closure of the study, the investigator or the head of the medical institution (where applicable) must maintain all site study records (except for those required by local regulations to be maintained elsewhere), in a safe and secure location.
- The records must be maintained to allow easy and timely retrieval, when needed (e.g., for a GSK audit or regulatory inspection) and must be available for review in conjunction with assessment of the facility, supporting systems, and relevant site staff.
- Where permitted by local laws/regulations or institutional policy, some or all of these records can be maintained in a format other than hard copy (e.g., microfiche, scanned, electronic); however, caution needs to be exercised before such action is taken.
- The investigator must ensure that all reproductions are legible and are a true and accurate copy of the original and meet accessibility and retrieval standards, including re-generating a hard copy, if required. Furthermore, the investigator must ensure there is an acceptable back-up of these reproductions and that an acceptable quality control process exists for making these reproductions.
- GSK will inform the investigator of the time period for retaining these records to comply with all applicable regulatory requirements. The minimum retention time will meet the strictest standard applicable to that site for the study, as dictated by any institutional requirements or local laws or regulations, GSK standards/procedures, and/or institutional requirements.
- The investigator must notify GSK of any changes in the archival arrangements, including, but not limited to, archival at an off-site facility or transfer of ownership of the records in the event the investigator is no longer associated with the site.

# 10.7. Provision of Study Results to Investigators, Posting of Information on Publically Available Clinical Trials Registers and Publication

Where required by applicable regulatory requirements, an investigator signatory will be identified for the approval of the clinical study report. The investigator will be provided reasonable access to statistical tables, figures, and relevant reports and will have the opportunity to review the complete study results at a GSK site or other mutually-agreeable location.

GSK will also provide the investigator with the full summary of the study results. The investigator is encouraged to share the summary results with the study subjects, as appropriate.

GSK will also provide the investigator with the randomization numbers assigned to the subjects of his/her study site after the completion of all analyses.

The procedures and timing for public disclosure of the results summary and for development of a manuscript for publication will be in accordance with GSK Policy.

# 10.8. Study Period

See Exhibit 1

#### 10.9. Study Administrative Structure

Sponsor information is included in Exhibit 2. List of Medical Institutions and Investigators is included in Exhibit 3.

#### 11. REFERENCES

Akizawa T, Makino H, Matsuo S, et al. Management of anemia in chronic kidney disease patients: baseline findings from Chronic Kidney Disease Japan Cohort Study. Clin Exp Nephrol. 2011;15:248-57.

Szczech LA, Barnhart HX., Inrig JK., et al. Secondary analysis of the CHOIR trial epoetin- $\alpha$  dose and achieved hemoglobin outcomes. Kidney International. 2008;74:791-8.

Guidelines for Renal Anemia in Chronic Kidney Disease issued by the Japanese Society for Dialysis Therapy in 2015. Journal of Japanese Society for Dialysis Therapy. 2016;49(2):89-158

MIRCERA. Product information in Europe (methoxy polyethylene glycol-epoetin beta). 2012-May. 2012.

KDIGO. KDIGO Clinical Practice Guideline for Anemia in Chronic Kidney Disease. Kidney International Supplement. 2012 Aug;2(4): 279-335.

# 12. APPENDICES

# 12.1. Appendix 1: Abbreviations and Trademarks

# **Abbreviations**

| ALT | Alanine Aminotransferase |
|---------------|----------------------------------------------------------|
| AST | Aspartate Aminotransferase |
| AUC | Area Under Curve |
| CKD | Chronic Kidney Disease |
| Cmax | Maximum concentration |
| СРК | Creatine Phosphokinase |
| CYP | Cytochrome P450 |
| DNA | Deoxyribonucleic Acid |
| EPO | Erythropoietin |
| EQ-5D-5L | EuroQol EuroQol 5 Dimension 5 Level Health Utility Index |
| EQ-VAS | EuroQol Visual Analogue Scale |
| ESA | Erythropoiesis-Stimulating Agent |
| FDA | Food and Drug Administration |
| FSH | Follicle Stimulating Hormone |
| GCP | Good Clinical Practice |
| GSK | GlaxoSmithKline |
| hCG | Human Chorionic Gonadotrophin |
| HD | Hemodialysis |
| HDL | High Density Lipoprotein |
| HDF | Hemodiafiltration |
| Hgb | Hemoglobin |
| HIF | Hypoxia-Inducible Factor |
| HRQoL | Health Related Quality of Life |
| HRT | Hormone Replacement Therapy |
| ICH | International Conference on Harmonization |
| INR | International Normalized Ratio |
| iPTH | Intact Parathyroid Hormone |
| ITT | Intent-to-Treat |
| IWRS | Interactive Web Recognition System |
| LDH | Lactate Dehydrogenase |
| LDL | Low Density Lipoprotein |
| MCS | Mental Component Summary |
| MCH | Mean Corpuscular Hemoglobin |
| MCHC | Mean Corpuscular Hemoglobin Concentration |
| MCV | Mean Corpuscular Volume |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | modified Intent-to-Treat |
| NYHA | New York Heart Association |
| PAH | Pulmonary Artery Hypertension |
| PCS | Physical Component Summary |
| PD | Peritoneal Dialysis |
| PHI | Prolyl Hydroxylase Inhibitor |
| PK | Pharmacokinetic |
| PP | Per-Protocol |
| PRO | Patient Reported Outcome |
| QT Interval | Q-T Interval |
| × 1 11101 vai | X 1 111041 1 m |

# **CONFIDENTIAL**

PHI201754

| QTc Interval | Q-T Interval Corrected for Heart Rate |
|--------------|---------------------------------------|
| QTcB | Bazett's Correction of QT Interval |
| RAP | Reporting and Analysis Plan |
| RDW | Red Blood Cell Distribution Width |
| RNA | Ribonucleic Acid |
| rhEPO | Recombinant human erythropoietin |
| SAE | Serious Adverse Event |
| sPAP | Systolic Pulmonary Artery Pressure |
| SRM | Study Reference Manual |
| TIBC | Total Iron Binding Capacity |
| TSAT | Transferrin Saturation |
| UIBC | Unsaturated iron Binding Capacity |
| VAS | Visual Analog Scale |
| VEGF | Vascular Endothelial Growth Factor |

# **Trademark Information**

| Trademarks of the GlaxoSmithKline group of companies |
|------------------------------------------------------|
| None |

| Trademarks not owned by the GlaxoSmithKline |
|---------------------------------------------|
| group of companies |
| Hemocue |
| Nesp® |

# 12.2. Appendix 2: Risk Assessment

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Daprodustat | | |
| Excessive erythropoiesis (polycythemia) leading to thrombosis and/or tissue ischemia | In animal studies, excessive erythropoiesis attributed to daprodustat was associated with vascular congestion, microthrombi, and tissue ischemia in a number of organs. Following review of clinical data received to date, this has not been identified as a safety concern for daprodustat. Phase 2 dose-ranging studies, and associated statistical and exposure response modelling has informed Phase 3 dose rationale, starting doses, dose levels, and dose adjustment scheme to optimize Hgb management. | <ul> <li>Specific eligibility criteria related to requirements for entry Hgb are detailed in Section 5.1.</li> <li>Hgb will be closely monitored throughout the dosing period as outlined in the Time and Events Table Section 7.1.</li> <li>Specific guidance for dose adjustment, dose interruption, or discontinuation of daprodustat based on achieved Hgb is provided in Section 6.4.1.</li> <li>These risks have been identified as AEs of special interest and will be monitored instreamly by the internal safety review team throughout the study period.</li> </ul> |
| Death, MI, stroke, heart failure, thromboembolic events, thrombosis of vascular access at Hgb levels which are within the normal range (i.e. not polycythemic conditions) | Marketed rhEPO/ESAs have been associated with an increased risk for death and serious cardiovascular events when used in patients with anemia of CKD. Following review of clinical data received to date, this has not been identified as a safety concern for daprodustat. | <ul> <li>Specific eligibility criteria related to CV risk are outlined in Section 5.2.</li> <li>Hgb will be closely monitored throughout the dosing period as outlined in the Time and Events Table Section 7.1.</li> <li>These risks have been identified as AEs</li> </ul> |

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Esophageal and gastric erosions Cancer-related mortality, tumor progression and recurrence | In animal studies, undesirable GI effects including emesis, abnormal feces and/or decreased food consumption/body weight loss and stomach erosions/ ulcers with hemorrhage were observed. In rodents stomach erosions observed with intravenous and oral administration of daprodustat. Gender-averaged systemic exposure (AUC) at the no observed adverse effect levels (NOAEL) are 3.3 -fold (monkeys) and 737 -fold (rats) above human exposure (25 mg). In clinical trials to date, mild-moderate GI signs and symptoms represent the most frequently reported adverse event, however causal association has not been established. Following review of clinical data received to date, GI erosions have not been identified as a safety concern for daprodustat. In clinical trials, use of rhEPO in patients with cancer has been associated with increased risk of cancer related morbidity and mortality. Administration of 60 mg/kg daprodustat to mice caused minimal increases in circulating VEGF while significant EPO increases were observed. In clinical studies up to 4 weeks duration, a dose-ordered increase in VEGF plasma concentrations, an angiogenic factor that has been implicated in tumor growth, was observed at doses ranging from 10 to | of special interest and will be monitored instreamly by the internal safety review team throughout the study period. Suspected Gl bleeding or significant symptoms consistent with erosion should be investigated diagnostically (i.e. endoscopic examination) as clinically warranted These risks have been identified as AEs of special interest and will be monitored instreamly by the internal safety review team throughout the study period. Specific eligibility criteria related to personal history of malignancy are outlined in Section 5.2 Stopping criteria for subjects with treatment emergent malignancy are outlined in Section 5.4. These risks have been identified as AEs of special interest and will be |
| | 150 mg. In clinical studies up to 24 weeks duration at doses up to 25 mg, changes in VEGF plasma concentrations were variable but similar relative to control. Following review of clinical data received to date, this has not been identified as a safety concern for daprodustat. | monitored instreamly by the internal safety review team throughout the study period. |
| Pulmonary artery hypertension (PAH) | A role for HIF-regulated pathways in the pathophysiology of PAH has been suggested based on well established effects of acute and chronic hypoxia in | These risks have been identified as AEs of special interest and will be monitored instreamly by the |

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| | man on the pulmonary vasculature (vasoconstriction), and by findings in patients with naturally occurring mutations that result in decreased HIF degradation (Smith, 2006; Formenti, 2011). | internal safety review team throughout the study period. |
| | There have been no histopathologic findings suggestive of PAH in pre-clinical safety studies (up to 13-weeks duration in mice and dog, up to 26-weeks in rat, and up to 39-weeks in monkeys. | |
| | Acute hypoxic challenge (rats): daprodustatA produced increases in peak right ventricular pressure (PRVP) during acute hypoxia that were slightly higher than the vehicle control group. These hypoxia-induced PRVP changes fall within the range of PRVP differences noted among non-treated rats. | |
| | Results from a clinical study of acute hypoxic challenge in healthy volunteers demonstrated that short-term therapy with daprodustat 5 mg or 100 mg has no clinically significant effect on echocardiographically estimated pulmonary artery systolic pressure (PASP) under either normoxic or hypoxic conditions. | |
| | ECHO assessments performed in Phase 2b studies (24 weeks treatment duration) did not identify any clinically meaningful changes in sPAP in subjects not on dialysis. In hemodialysis subjects, mean absolute change from baseline in sPAP was similar for both treatment groups; however, there was a numeric imbalance (GSK Total: 8 [7%]; Control 0) in subjects reaching the sPAP PCI (>20 mmHg increase from baseline). Regarding this imbalance, there were a number of confounding factors in the study, most notably a 4.5:1 randomization scheme and inconsistency in timing of ECHOs relative to dialysis day. Additionally, 2 of 3 subjects with resolution of sPAP on safety follow-up ECHOs had confounding conditions that could contribute to resolution other than discontinuation of study treatment; and there was no dose relationship for subjects meeting the sPAP PCI criterion. Overall, there is insufficient evidence to conclude a relationship to treatment with daprodustat. | |
| | Following review of clinical data received to date, this has not been identified as a safety concern for daprodustat. | |
| Cardiomyopathy | Published data suggest that cardiac effects of HIF stabilization are likely a function of the mechanism, extent, and duration of the effects, and can range from protective to detrimental depending upon the specific model and experimental conditions utilized. | These risks have been identified as AEs of special interest and will be monitored instreamly by the internal safety review team throughout the study |

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Proliferative retinopathy, macular edema, choroidal neovascularization | Small increases in cardiac troponin in 6 month rat study were consistent with the background finding of spontaneous rodent cardiomyopathy. There were no elevations observed in cardiac troponin in 9 month monkey study. Cardiomyopathy has not been associated with naturally occurring mutation in man which results in increased HIF stabilization. ECHO assessments performed in phase 2b studies (24 weeks treatment duration) did not identify any clinically meaningful changes in LVEF. Following review of clinical data received to date, this has not been identified as a safety concern for daprodustat. Increases in local (ocular) VEGF production with retinal neovascularization and macular edema observed in diabetic retinopathy and to choroidal leakage, edema and neovascularization seen in age-related macular degeneration (Campochiaro, 2006). Administration of 60 mg/kg daprodustat to mice caused minimal increases in circulating VEGF while significant EPO increases were observed. No ocular abnormalities were seen in non-clinical studies of up to 13 weeks duration in mice and dogs, 26 weeks in rats, and 39-weeks in monkeys. In clinical studies up to 4 weeks duration, a dose-ordered increase in VEGF plasma concentrations was observed at doses ranging from 10 to 150 mg. In studies up to 24 weeks duration at doses up to 25 mg, changes in VEGF plasma concentrations were variable but similar relative to control. Ophthalmologic assessments performed in phase 2b studies (24 weeks treatment duration) did not identify any clinically meaningful changes in proliferative retinopathy, macular | <ul> <li>Ophthalmology exams will be performed during screening, at approximately Week 12 on-study, and at the end of treatment.</li> <li>These risks have been identified as AEs of special interest and will be monitored instreamly by the internal safety review team throughout the study period.</li> <li>Suspected proliferative retinopathy, macular edema, choroidal neovascularization or symptoms consistent with these events should be investigated by ophthalmologic consultation as clinically warranted.</li> </ul> |
| | edema, or choroidal neovascularization. Following review of clinical data received to date, this has not been identified as a safety concern for daprodustat. | |
| Exacerbation of rheumatoid arthritis | In inflamed rheumatic joints, activation of HIF- related genes | These risks have been identified as AEs of special |

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| | secondary to decreased oxygen and pro-inflammatory cytokines has been postulated to contribute to the neo-angiogenesis, proliferation and infiltration of rheumatoid synovial fibroblasts (Westra, 2010; Muz, 2009). No abnormalities seen in non-clinical studies conducted to date. Following review of clinical data received to date, this has not been identified as a safety concern for daprodustat. | interest and will be monitored instreamly by the internal safety review team throughout the study period. |
| Orug-drug interactions | Co-administration of daprodustat with a strong CYP2C8 inhibitor increased the Cmax and AUC of daprodustat, 4- and 19-fold, respectively, while co-administration of a weak inhibitor increased the Cmax and AUC of daprodustat by 1.3- and 1.5-fold, respectively. Population PK analysis from completed Phase 2 studies suggests that co-administration of daprodustat with a moderate CYP2C8 inhibitor, leads to a $\sim$ 2-fold increase in AUC, with no clinically-significant increase in the measured Hgb response. Daprodustat is an inhibitor of CYP2C8 in vitro, with an IC50 value of 21 $\mu$ M. Population PK analysis from completed Phase 2 studies suggests that co-administration of daprodustat with clopidogrel (a moderate CYP2C8 inhibitor) leads to a $\sim$ 2-fold increase in AUC, with no clinically-significant increase in the measured Hgb response. Co-administration of daprodustat with moderate CYP2C8 inhibitors (i.e., clopidogrel, teriflunomide, deferasirox) should be performed with caution. Co-administration of daprodustat with potent BCRP inhibitors has the potential to increase exposure of daprodustat. Use of BCRP inhibitors (mostly weak) was found to result in a small change in metabolite exposure (20% increase in AUC). Daprodustat is an inhibitor of OATP1B1/1B3 in vitro, with IC50 values of 6 $\mu$ M and 11 $\mu$ M, respectively. A clinical drug interaction study between 25mg daprodustat with either a CYP2C8 substrate or an OATP1B1/1B3 substrate showed that there is no PK interaction at this dose of daprodustat. | Co-administration of daprodustat with strong CYP2C8 inhibitors (e.g., gemfibrozil) and inducers (e.g., rifampin/rifampicin) is not permitted as outlined in Section 6.11.2. Co-administration of daprodustat with moderate CYP2C8 inhibitors (i.e., clopidogrel, teriflunomide, deferasirox) should be performed with caution. Specific guidance on the management of potential drug-drug interactions and concomitant medications is provided in Section 6.11. Hgb will be closely monitored throughout the dosing period as outlined in the Time and Events Table Section 7.1. Specific guidance for dose adjustment, dose interruption, or discontinuation of daprodustat based on achieved Hgb is provided in Section 6.4.1. Safety data will be monitored instreamly by the internal safety review team throughout the study period. |
| Other | | |
| SA risks (Control) | See risks outlined in table for daprodustat for Excessive erythropoiesis | The same mitigation strategies have been indentified |

2015N266251\_02 **CONFIDENTIAL** PHI201754

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| | (polycythemia) leading to thrombosis and/or tissue ischemia; Risk of | in acoordance with the mitigation strategies for |
| | MI, stroke, thromboembolic events, thrombosis of vascular access; and | daprodustat |
| | risk of cancer-related mortality and tumor progression. | Monitor instreamly blood pressure throughout |
| | | the study as scheduled in Table 10. |
| | Uncontrolled hypertension. | Specific eligibility criteria related to personal |
| | | history of pure red cell aplasia are outlined in |
| | Pure red cell aplasia | Section 5.2. |
| | | Liver function will be monitored throughout |
| | Hepatic function disorder with increase of ALT and Gamma- | the dosing period as outlined in the Time and |
| | glutamyltransferase, and jaundice have been reported as adverse | Events Table provided in Section 7.1. |
| | drug reactions according to the prescribing information of | Î |
| | darbepoetin alfa. | |

#### References

Campochiaro PA and the First ARVO/Pfizer Institute Working Group. Ocular versus Extraocular Neovascularization: Mirror Images or Vague Resemblances. Invest Ophthalmol & Vis Sci. 2006;47:462-74.

Formenti F, Beer PA, Croft QP, et al. Cardiopulmonary function in two human disorders of the hypoxia-inducible factor (HIF) pathway: von Hippel-Lindau disease and HIF-2alpha gain-of-function mutation. FASEB J. 2011;25(6):2001-11.

Muz B, Khan MN, Kiriakidis S, et al. Hypoxia. The role of hypoxia and HIF-dependent signalling events in rheumatoid arthritis. Arthritis Research & Therapy. 2009;11:201.

Smith TG, Brooks JT, Balanos GM, et al. Mutation of von Hippel-Lindau Tumour Suppressor and Human Cardiopulmonary Physiology . PLoS Med. 2006;3:1178-86.

Westra J, Molema G and Kallenberg CG. Hypoxia-Inducible Factor-1 as Regulator of Angiogenesis in Rheumatoid Arthritis - Therapeutic Implications. Current Medicinal Chemistry 2010;17(3):254-63.

# 12.3. Appendix 3: Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of reproductive potential

This list does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis.

- 1. Contraceptive subdermal implant that meets the Prescribing Information effectiveness criteria including a <1% rate of failure per year, as stated in the Prescribing Information
- 2. Intrauterine device or intrauterine system that meets the Prescribing Information effectiveness criteria including a <1% rate of failure per year, as stated in the Prescribing Information [Hatcher, 2011]
- 3. Combined estrogen and progestogen oral contraceptive [Hatcher, 2011]
- 4. Injectable progestogen [Hatcher, 2011]
- 5. Contraceptive vaginal ring [Hatcher, 2011]
- 6. Percutaneous contraceptive patches [Hatcher, 2011]
- 7. Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject [Hatcher, 2011].

These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the Prescribing Information. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

#### References

Trussell J, Contraceptive Efficacy. In: Hatcher RA, Trussell J, Nelson AL, Cates W, Kowal D, and Policar M (editors). Contraceptive Technology: Twentieth Revised Edition. New York: Ardent Media, 2011.

## 12.4. Appendix 4: Collection of Pregnancy Information

- Investigator will collect pregnancy information on any female subject, who becomes pregnant while participating in this study
- Information will be recorded on the appropriate form and submitted to GSK within 2 weeks of learning of a subject's pregnancy.
- Subject will be followed to determine the outcome of the pregnancy. The investigator will collect follow up information on mother and infant, which will be forwarded to GSK. Generally, follow-up will not be required for longer than 6 to 8 weeks beyond the estimated delivery date.
- Any termination of pregnancy will be reported, regardless of fetal status (presence or absence of anomalies) or indication for procedure.
- While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or elective termination of a pregnancy will be reported as an AE or SAE.
- A spontaneous abortion is always considered to be an SAE and will be reported as such.
- Any SAE occurring as a result of a post-study pregnancy which is considered reasonably related
  to the study treatment by the investigator, will be reported to GSK as described in Section 12.6.
   Appendix 6. While the investigator is not obligated to actively seek this information in former
  study participants, he or she may learn of an SAE through spontaneous reporting.

#### Any female subject who becomes pregnant while participating

• will discontinue study medication or be withdrawn from the study

# 12.5. Appendix 5: Liver Safety Required Actions and Follow up Assessments Phase III-IV liver chemistry stopping and increased monitoring criteria have been designed to assure subject safety and evaluate liver event etiology (in alignment with the FDA premarketing clinical liver safety guidance).

Phase III-IV liver chemistry stopping criteria and required follow up assessments

| Liver Chemistr | Liver Chemistry Stopping Criteria - Liver Stopping Event | |
|---|---|---|
| ALT-absolute | ALT ≥ 8xULN | |
| ALT Increase | $ALT \ge 5xULN$ but $\le 8xULN$ persists for $\ge 2$ weeks | |
| | ALT $\geq$ 3xULN but $\leq$ 5xULN persists for $\geq$ 4 weeks | |
| Bilirubin <sup>1, 2</sup> | ALT $\geq$ 3xULN and bilirubin $\geq$ 2xULN (>35% direct bilirubin) | |
| INR <sup>2</sup> | ALT $\geq$ 3xULN and INR>1.5, if INR measured | |
| Cannot | ALT $\geq$ 5xULN but $\leq$ 8xULN and cannot be monitored weekly for $\geq$ 2 weeks | |
| Monitor | ALT $\geq$ 3xULN but $\leq$ 5xULN and cannot be monitored weekly for $\geq$ 4 weeks | |
| Symptomatic <sup>3</sup> | ALT $\geq$ 3xULN associated with symptoms (new or worsening) believed to be related | |
| Required Action | liver injury or hypersensitivity ns and Follow up Assessments follow | wing ANY Liver Stopping Event |
| Actions | | Follow Up Assessments |
| • Immediate | ly discontinue study treatment | Viral hepatitis serology <sup>4</sup> |
| • Report the | event to GSK within 24 hours | Only in those with underlying chronic |
| • Complete | the liver event CRF and complete | hepatitis B at study entry (identified by |
| an SAE da | ta collection tool if the event also | positive hepatitis B surface antigen) and |
| meets the | criteria for an SAE <sup>2</sup> | quantitative hepatitis B DNA |
| • Perform liver event follow up assessments | | Blood sample for pharmacokinetic (PK) |
| Monitor the subject until liver chemistries | | analysis, obtained within 24 hours after las |
| | abilize, or return to within baseline | dose <sup>5</sup> |
| | ITORING below) | • Serum creatine phosphokinase (CPK) and |
| Do not restart/rechallenge subject with | | lactate dehydrogenase (LDH). |
| study treatment unless allowed per protocol | | • Fractionate bilirubin, if total |
| = | Medical Governance approval <b>is</b> | bilirubin≥2xULN |
| granted | | Obtain complete blood count with |
| • If restart/re | echallenge <b>not allowed or not</b> | differential to assess eosinophilia |
| granted, permanently discontinue study | | Record the appearance or worsening of |
| treatment and may continue subject in the | | clinical symptoms of liver injury, or |
| study for any protocol specified follow up | | hypersensitivity, on the AE report form |
| assessments | | Record use of concomitant medications on |
| • | | the concomitant medications report form |
| MONITORING: | | including acetaminophen, herbal remedies. |
| | r INR criteria: | other |
| Repeat liver chemistries (include ALT, AST, | | • over the counter medications. |
| alkaline phosphatase, bilirubin) and perform | | Record alcohol use on the liver event |

# liver event follow up assessments within 24 hrs

- Monitor subjects twice weekly until liver chemistries resolve, stabilize or return to within baseline
- A specialist or hepatology consultation is recommended

#### For All other criteria:

- Repeat liver chemistries (include ALT, AST, alkaline phosphatase, bilirubin) and perform liver event follow up assessments within
   24-72 hrs
- Monitor subjects weekly until liver chemistries resolve, stabilize or return to within baseline

alcohol intake case report form

#### For bilirubin or INR criteria:

- Anti-nuclear antibody, anti-smooth muscle antibody, Type 1 anti-liver kidney microsomal antibodies, and quantitative total immunoglobulin G (IgG or gamma globulins).
- Serum acetaminophen adduct HPLC assay (quantifies potential acetaminophen contribution to liver injury in subjects with definite or likely acetaminophen use in the preceding week [James, 2009]).
- Liver imaging (ultrasound, magnetic resonance, or computerised tomography) and /or liver biopsy to evaluate liver disease; complete Liver Imaging and/or Liver Biopsy CRF forms.
- 1. Serum bilirubin fractionation should be performed if testing is available. If serum bilirubin fractionation is not immediately available, discontinue study treatment for that subject if  $ALT \ge 3xULN$  and bilirubin  $\ge 2xULN$ .
- 2. All events of ALT ≥ 3xULN and bilirubin ≥ 2xULN (>35% direct bilirubin) or ALT ≥ 3xULN and INR>1.5, if INR measured which may indicate severe liver injury (possible 'Hy's Law'), must be reported as an SAE (excluding studies of hepatic impairment or cirrhosis); INR measurement is not required and the threshold value stated will not apply to subjects receiving anticoagulants
- New or worsening symptoms believed to be related to liver injury (such as fatigue, nausea, vomiting, right upper quadrant pain or tenderness, or jaundice) or believed to be related to hypersensitivity (such as fever, rash or eosinophilia)
- 4. Includes: Hepatitis A IgM antibody; Hepatitis B surface antigen and Hepatitis B Core Antibody (IgM); Hepatitis C RNA; Cytomegalovirus IgM antibody; Epstein-Barr viral capsid antigen IgM antibody (or if unavailable, obtain heterophile antibody or monospot testing); Hepatitis E IgM antibody or Hepatitis E RNA
- 5. PK sample may not be required for subjects known to be receiving placebo or non-GSK comparator treatments. Record the date/time of the PK blood sample draw and the date/time of the last dose of study treatment prior to blood sample draw on the CRF. If the date or time of the last dose is unclear, provide the subject's best approximation. If the date/time of the last dose cannot be approximated OR a PK sample cannot be collected in the time period indicated above, do not obtain a PK sample. Instructions for sample handling and shipping are in the SRM.

#### Phase III-IV liver chemistry increased monitoring criteria with continued therapy

| Liver Chemistry Increased Monitoring Criteria – Liver Monitoring Event | |
|---|---|
| Criteria | Actions |
| ALT ≥5xULN and <8xULN and bilirubin <2xULN without symptoms believed to be related to liver injury or hypersensitivity, and who can be monitored weekly for 2 weeks. OR | <ul> <li>Notify the GSK medical monitor within 24 hours of learning of the abnormality to discuss subject safety.</li> <li>Subject can continue study treatment</li> <li>Subject must return weekly for repeat liver</li> </ul> |

ALT  $\ge 3$ xULN and < 5xULN and bilirubin < 2xULN without symptoms believed to be related to liver injury or hypersensitivity, and who can be monitored weekly for 4 weeks.

- chemistries (ALT, AST, alkaline phosphatase, bilirubin) until they resolve, stabilise or return to within baseline
- If at any time subject meets the liver chemistry stopping criteria, proceed as described above
- If ALT decreases from ALT ≥5xULN and <8xULN to ≥3xULN but <5xULN, continue to monitor liver chemistries weekly.
- If, after 4 weeks of monitoring, ALT <3xULN and bilirubin <2xULN, monitor subjects twice monthly until liver chemistries normalize or return to within baseline.

#### References

James LP, Letzig L, Simpson PM, et al. Pharmacokinetics of Acetaminophen-Protein Adductsin Adults with Acetaminophen Overdose and Acute Liver Failure. Drug Metab Dispos. 2009;37:1779-84.

# 12.6. Appendix 6: Definition of and Procedures for Recording, Evaluating, Follow-Up and Reporting of Adverse Events

#### 12.6.1. Definition of Adverse Events

#### **Adverse Event Definition:**

- An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
- NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.

#### Events meeting AE definition include:

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or other safety assessments (e.g., ECGs, radiological scans, vital signs measurements), including those that worsen from baseline, and felt to be clinically significant in the medical and scientific judgement of the investigator.
- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after study treatment administration even though it may have been present prior to the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study treatment or a
  concomitant medication (overdose per se will not be reported as an AE/SAE unless this is an
  intentional overdose taken with possible suicidal/self-harming intent. This should be reported
  regardless of sequelae).
- "Lack of efficacy" or "failure of expected pharmacological action" per se will not be reported as an AE or SAE. However, the signs and symptoms and/or clinical sequelae resulting from lack of efficacy will be reported if they fulfil the definition of an AE or SAE.

#### Events **NOT** meeting definition of an AE include:

- Any clinically significant abnormal laboratory findings or other abnormal safety assessments
  which are associated with the underlying disease, unless judged by the investigator to be more
  severe than expected for the subject's condition.
- The disease/disorder being studied or expected progression, signs, or symptoms of the disease/disorder being studied, unless more severe than expected for the subject's condition.
- Medical or surgical procedure (e.g., endoscopy, appendectomy): the condition that leads to the procedure is an AE.
- Situations where an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).
- Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen.

#### 12.6.2. Definition of Serious Adverse Events

If an event is not an AE per definition above, then it cannot be an SAE even if serious conditions are met (e.g., hospitalization for signs/symptoms of the disease under study, death due to progression of disease, etc).

#### Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose:

#### a. Results in death

#### b. Is life-threatening

#### NOTE:

The term 'life-threatening' in the definition of 'serious' refers to an event in which the subject was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.

# c. Requires hospitalization or prolongation of existing hospitalization

#### NOTE:

- In general, hospitalization signifies that the subject has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or out-patient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious.
- Hospitalization for elective treatment of a pre-existing condition that did not worsen from baseline is not considered an AE.

#### d. Results in disability/incapacity

#### NOTE:

- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (e.g. sprained ankle) which may interfere or prevent everyday life functions but do not constitute a substantial disruption

# e. Is a congenital anomaly/birth defect

#### f. Other situations:

- Medical or scientific judgment should be exercised in deciding whether reporting is appropriate
  in other situations, such as important medical events that may not be immediately life-threatening
  or result in death or hospitalization but may jeopardize the subject or may require medical or
  surgical intervention to prevent one of the other outcomes listed in the above definition. These
  should also be considered serious.
- Examples of such events are invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse

#### g. Is associated with liver injury and impaired liver function defined as:

- ALT  $\geq$  3xULN and total bilirubin\*  $\geq$  2xULN (>35% direct), or
- ALT  $\geq 3$ xULN and INR\*\* > 1.5.

- \* Serum bilirubin fractionation should be performed if testing is available; (for ND patients only) if unavailable, record presence of detectable urinary bilirubin on dipstick, indicating direct bilirubin elevations and suggesting liver injury. If fractionation is unavailable and ALT  $\geq$  3xULN and total bilirubin  $\geq$  2xULN, then the event is still to be reported as an SAE.
- \*\* INR testing not required per protocol and the threshold value does not apply to subjects receiving anticoagulants. If INR measurement is obtained, the value is to be recorded on the SAE form.

#### 12.6.3. Definition of Cardiovascular Events

# Cardiovascular Events (CV) Definition:

Investigators will be required to fill out the specific CV event page of the CRF for the following AEs and SAEs:

- Myocardial infarction/unstable angina
- Congestive heart failure
- Arrhythmias
- Valvulopathy
- Pulmonary hypertension
- Cerebrovascular events/stroke and transient ischemic attack
- Peripheral arterial thromboembolism
- Deep venous thrombosis/pulmonary embolism
- Revascularization

#### 12.6.4. Recording of AEs and SAEs

#### **AEs and SAE Recording:**

- When an AE/SAE occurs, it is the responsibility of the investigator to review all documentation (e.g., hospital progress notes, laboratory, and diagnostics reports) relative to the event.
- The investigator will then record all relevant information regarding an AE/SAE in the CRF
- It is not acceptable for the investigator to send photocopies of the subject's medical records to GSK in lieu of completion of the GSK, AE/SAE CRF page.
- There may be instances when copies of medical records for certain cases are requested by GSK.
   In this instance, all subject identifiers, with the exception of the subject number, will be blinded on the copies of the medical records prior to submission of to GSK.
- The investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. In such cases, the diagnosis will be documented as the AE/SAE and not the individual signs/symptoms.
- PRO questionnaires and the collection of AE data are independent components of the study.
- Responses to each question in PRO questionnaire will be treated in accordance with standard scoring and statistical procedures detailed by the scale's developer.
- The use of a single question from a multidimensional health survey to designate a cause-effect relationship to an AE is inappropriate.

#### 12.6.5. Evaluating AEs and SAEs

#### **Assessment of Intensity**

The investigator will make an assessment of intensity for each AE and SAE reported during the study and will assign it to one of the following categories:

- Mild: An event that is easily tolerated by the subject, causing minimal discomfort and not interfering with everyday activities.
- Moderate: An event that is sufficiently discomforting to interfere with normal everyday activities
- Severe: An event that prevents normal everyday activities. an AE that is assessed as severe will not be confused with an SAE. Severity is a category utilized for rating the intensity of an event; and both AEs and SAEs can be assessed as severe.
- An event is defined as 'serious' when it meets at least one of the pre-defined outcomes as described in the definition of an SAE.

#### **Assessment of Causality**

- The investigator is obligated to assess the relationship between study treatment and the occurrence of each AE/SAE.
- A "reasonable possibility" is meant to convey that there are facts/evidence or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- The investigator will use clinical judgment to determine the relationship.
- Alternative causes, such as natural history of the underlying diseases, concomitant therapy, other
  risk factors, and the temporal relationship of the event to the study treatment will be considered
  and investigated.
- The investigator will also consult the Investigator Brochure (IB) and/or Product Information, for marketed products, in the determination of his/her assessment.
- For each AE/SAE the investigator <u>must</u> document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.
- There may be situations when an SAE has occurred and the investigator has minimal information to include in the initial report to GSK. However, it is very important that the investigator always make an assessment of causality for every event prior to the initial transmission of the SAE data to GSK.
- The investigator may change his/her opinion of causality in light of follow-up information, amending the SAE data collection tool accordingly.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.

#### Follow-up of AEs and SAEs

- The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as may be indicated or as requested by GSK to elucidate as fully as possible the nature and/or causality of the AE or SAE.
- The investigator is obligated to assist. This may include additional laboratory tests or investigations, histopathological examinations or consultation with other health care
- professionals.
- If a subject dies during participation in the study or during a recognized follow-up period, the investigator will provide GSK with a copy of any post-mortem findings, including histopathology.
- New or updated information will be recorded in the originally completed CRF.
- The investigator will submit any updated SAE data to GSK within the designated reporting time frames.

#### 12.6.6. Reporting of SAEs to GSK

#### SAE reporting to GSK via electronic data collection tool

- Primary mechanism for reporting SAEs to GSK will be the electronic data collection tool
- If the electronic system is unavailable for greater than 24 hours, the site will use the paper SAE data collection tool and fax it to the SAE contact.
- Site will enter the serious adverse event data into the electronic system as soon as it becomes available.
- The investigator (or subinvestiagtor) will mark a check against 'reviewed' box in the lower part of the eCRF page within 72 hours after reporting of SAE to ensure that the causality of AE has been reviewed.
- After the study is completed at a given site, the electronic data collection tool (e.g., InForm system) will be taken off-line to prevent the entry of new data or changes to existing data
- If a site receives a report of a new SAE from a study subject or receives updated data on a previously reported SAE after the electronic data collection tool has been taken off-line, the site can report this information on a paper SAE form or to the SAE contact by telephone.
- Contacts for SAE receipt can be found at the beginning of this protocol on the Sponsor/Medical Monitor Contact Information page.

### 12.7. Appendix 7 - Genetic Research Background

Naturally occurring genetic variation may contribute to inter-individual variability in response to medicines, as well as an individual's risk of developing specific diseases. Genetic factors associated with disease characteristics may also be associated with response to therapy, and could help to explain some clinical study outcomes. For example, genetic variants associated with age-related macular degeneration (AMD) are reported to account for much of the risk for the condition [Gorin, 2012] with certain variants reported to influence treatment response [Chen, 2012]. Thus, knowledge of the genetic etiology of disease may better inform understanding of disease and the development of medicines. Additionally, genetic variability may impact the pharmacokinetics (absorption, distribution, metabolism, and elimination), or pharmacodynamics (relationship between concentration and pharmacologic effects or the time course of pharmacologic effects) of a specific medicine and/or clinical outcomes (efficacy and/or safety) observed in a clinical study.

#### **Genetic Research Objectives and Analyses**

The objective of the genetic research is to understand the response to daprodustat. To achieve this objective, the relationship between genetic variants and the followings may be investigated.

- Response to medicine, including daprodustat, ESA, other study medicines or any concomitant medicines;
- Nephrogenic anemia and related conditions susceptibility, severity, and progression

•

Genetic data may be generated while the study is underway or following completion of the study. Genetic evaluations may include focused candidate gene approaches and/or examination of a large number of genetic variants throughout the genome (whole genome analyses). Genetic analyses which will be conducted for this study will utilize data collected in the study and will be limited to understanding the objectives highlighted above. Analyses may be performed using data from multiple clinical studies related to daprodustat to investigate these research objectives.

Appropriate descriptive and/or statistical analysis methods will be used. A detailed description of any planned analyses will be documented in a Reporting and Analysis Plan (RAP) prior to initiation of the analysis. Planned analyses and results of genetic investigations will be reported either as part of the clinical RAP and study report, or in a separate genetics RAP and report, as appropriate.

#### **Study Population**

Any subject who is enrolled in the study can participate in the genetic research. Any subject who has received an allogeneic bone marrow transplant must be excluded from the genetic research.

#### **Study Assessments and Procedures**

A key component of successful genetic research is the collection of samples during clinical studies. Collection of samples, even when no *a priori* hypothesis has been identified, may enable future genetic analyses to be conducted, align with the purpose of the genetic research, to help understand variability in disease and medicine response.

• A 6 mL blood sample will be taken for DNA extraction. A Blood sample is collected at the baseline visit, after the subject has been randomized and provided informed consent for genetic research. Instructions for collection and shipping of the genetic sample are described in the laboratory manual. The DNA from the blood sample may undergo quality control analyses to confirm the integrity of the sample. If there are concerns regarding the quality of the sample, then the sample may be destroyed. The blood sample is taken on a single occasion unless a duplicate sample is required due to an inability to utilize the original sample.

The genetic sample is labelled (or "coded") with the same study specific number used to label other samples and data in the study. This number can be traced or linked back to the subject by the investigator or site staff. Coded samples do not carry personal identifiers (such as name or social security number).

Samples will be stored securely and may be kept for up to 15 years after the last subject completes the study, or GSK may destroy the samples sooner. GSK or those working with GSK (for example, other researchers) will only use samples collected from the study for the purpose stated in this protocol and in the informed consent form. Samples may be used as part of the development of a companion diagnostic to support the GSK medicinal product.

Subjects can request their sample to be destroyed at any time.

#### **Informed Consent**

Subjects who do not wish to participate in the genetic research may still participate in the study. Genetic informed consent must be obtained prior to any blood being taken.

#### Subject Withdrawal from Study

If a subject who has consented to participate in genetic research withdraws from the clinical study for any reason other than being lost to follow-up, the subject will be given a choice of one of the following options concerning the genetic sample, if already collected:

- Continue to participate in the genetic research in which case the genetic DNA sample is retained
- Discontinue participation in the genetic research and destroy the genetic DNA sample

If a subject withdraws consent for genetic research or requests sample destruction for any reason, the investigator must complete the appropriate documentation to request sample destruction within the timeframe specified by GSK and maintain the documentation in the site study records.

Genotype data may be generated during the study or after completion of the study and may be analyzed during the study or stored for future analysis.

• If a subject withdraws consent for genetic research and genotype data has not been analyzed, it will not be analyzed or used for future research.

• Genetic data that has been analyzed at the time of withdrawn consent will continue to be stored and used, as appropriate.

•

#### Screen and Baseline Failures

If a sample for genetic research has been collected and it is determined that the subject does not meet the entry criteria for participation in the study, then the investigator should instruct the subject that their genetic sample will be destroyed. No forms are required to complete this process as it will be completed as part of the consent and sample reconciliation process. In this instance a sample destruction form will not be available to include in the site files.

#### Provision of Study Results and Confidentiality of Subject's Genetic Data

GSK may summarize the genetic research results in the clinical study report, or separately and may publish the results in scientific journals.

GSK may share genetic research data with other scientists to further scientific understanding in alignment with the informed consent. GSK does not inform the subject, family members, insurers, or employers of individual genotyping results that are not known to be relevant to the subject's medical care at the time of the study, unless required by law. This is due to the fact that the information generated from genetic studies is generally preliminary in nature, and therefore the significance and scientific validity of the results are undetermined. Further, data generated in a research laboratory may not meet regulatory requirements for inclusion in clinical care.

#### References

Chen H, Yu KD, Xu GZ. Association between Variant Y402H in Age-Related Macular Degeneration (AMD) Susceptibility Gene CFH and Treatment Response of AMD: A Meta-Analysis. PloS One 2012;7:e42464.

Gorin MB. Genetic insights into age-related macular degeneration: Controversies addressing risk, causality, and therapeutics. Mol. Aspects. Med. 2012;33:467-86.

#### 12.8. Appendix 8: Definition of and Procedures for Documenting Medical Device **Incidents**

#### 12.8.1. **Definitions of a Medical Device Incident**

The detection and documentation procedures described in this protocol apply to all medical devices provided for use in the study (see Section 6.2 for the list of the medical devices).

#### Medical Device Incident Definition:

- Incident Any malfunction or deterioration in the characteristics and/or performance of a device, as well as any inadequacy in the labeling or the instructions for use which, directly or indirectly, might lead to or might have led to the death of a patient/user/other persons or to a serious deterioration in their state of health.
- Not all incidents lead to death or serious deterioration in health. The non-occurrence of such a result might have been due to other fortunate circumstances or to the intervention of health care personnel.

#### It is sufficient that:

- an incident associated with a device happened and
- the incident was such that, if it occurred again, might lead to death or a serious deterioration in

A serious deterioration in state of health can include:

- life-threatening illness
- permanent impairment of body function or permanent damage to a body structure
- a condition necessitating medical or surgical intervention to prevent one of the above
- fetal distress, fetal death or any congenital abnormality or birth defects

#### Examples of incidents

- a patient, user, care giver or professional is injured as a result of a medical device failure or its
- a patient's treatment is interrupted or compromised by a medical device failure
- misdiagnosis due to medical device failure leads to inappropriate treatment
- a patient's health deteriorates due to medical device failure

#### 12.8.1.1. **Documenting Medical Device Incidents**

#### Medical Device Incident Documenting:

- Any medical device incident occurring during the study will be documented in the subject's medical records, in accordance with the investigator's normal clinical practice, and on the appropriate form.
- For incidents fulfilling the definition of an AE or an SAE, the appropriate AE/SAE CRF page will be completed as described in Appendix 6 (Section 12.6).
- The form will be completed as thoroughly as possible and signed by the investigator before

#### transmittal to GSK.

- It is very important that the investigator provides his/her assessment of causality to the medical device provided by GSK at the time of the initial report, and describes any corrective or remedial actions taken to prevent recurrence of the incident.
- A remedial action is any action other than routine maintenance or servicing of a device where such action is necessary to prevent recurrence of an incident. This includes any amendment to the design to prevent recurrence.

#### 12.9. Appendix 9: Protocol Changes

#### 12.9.1. Amendment 1 — Summary of Changes and Rationale

This is applicable to all study sites.

#### List of Protocol Changes with Rationale for Each

#### **Sponsor Signatory:**

#### **Original Text:**

Hiromu Nakajima

Head,

Medicines Development,

Japan Development and Medical Affairs (JDMA),

GlaxoSmithKline K. K.

#### **Revised Text:**

Kihito Takahashi

Director

Japan Development and Medical Affairs (JDMA),

GlaxoSmithKline K. K.

#### Reason:

To reflect change of Sponsor Signatory.

#### **Emergency Contact**

#### **Original Text:**

Emergency Contact at night and holiday (Mon to Fri 6pm to 10am, Sat, Sun, national holiday and year-end and New Year holidays)

Bell Medical Solutions Inc.

#### **Revised Text:**

Emergency Contact at night and holiday (Mon to Fri 6pm to 10am, Sat, Sun, national holiday and year-end and New Year holidays)

BI Medical Inc.

#### Reason:

To reflect change of company name.

#### **Exclusion Criteria**

#### **Original Text:**

- 8. Liver disease (if any of the following occurs):
  - ALT > 2 x upper limit of normal (ULN)

• Bilirubin > 1.5 x ULN (If bilirubin fractions are measured and direct bilirubin is < 35%, isolated bilirubin > 1.5 x ULN will be acceptable.)

#### **Revised Text:**

- 8. Liver disease (if any of the following occurs):
  - (Screening verification only): ALT > 2 x upper limit of normal (ULN)
  - (<u>Screening verification only</u>): Bilirubin > 1.5 x ULN (If bilirubin fractions are measured and direct bilirubin is < 35%, isolated bilirubin > 1.5 x ULN will be acceptable.)

#### Reason:

To clarify the timing of eligibility assessment regarding exclusion criteria.

#### 6.11.2. Prohibited Medications and Non-Drug Therapies

#### **Original Text:**

None

#### **Revised Text:**

Use of the following drug; during the treatment period:

• Erythropoietin (e.g., epoetin/ darbepoetin alfa/ epoetin beta pegol)

Note: excluding darbepoetin alfa (brand name: Nesp) supplied by GSK.

#### Reason:

To clarify that there is a limitation to use erythropoietin.

#### 7.1. Time and Events Table

#### **Original Text:**

Unless otherwise specified, all assessments should occur before dialysis on the day.

#### **Revised Text:**

<u>In any case, the study visit should occur on the first dialysis session day of the week.</u> Unless otherwise specified, all assessments should occur before dialysis on the day.

#### Reason:

To clarify study procedure.

#### 7.4.2. Adverse Events of Special Interest

#### **Original Text:**

• Thrombosis and/or tissue ischemia secondary to excessive erythropoiesis

- Death, myocardial infarction (MI), stroke, venous thromboembolism, thrombosis of vascular access
- Cardiomyopathy
- Pulmonary artery hypertension (PAH)
- Cancer-related mortality and tumor progression and recurrence
- Esophageal and gastric erosions
- Proliferative retinopathy, macular edema, choroidal neovascularization
- Exacerbation of <u>inflammatory joint disease (e.g., rheumatoid arthritis)</u>

#### **Revised Text:**

- Thrombosis and/or tissue ischemia secondary to excessive erythropoiesis
- Death, myocardial infarction (MI), stroke, <u>congestive heart failure</u>, venous thromboembolism, thrombosis of vascular access
- Cardiomyopathy
- Pulmonary artery hypertension (PAH)
- Cancer-related mortality and tumor progression and recurrence
- Esophageal and gastric erosions
- Proliferative retinopathy, macular edema, choroidal neovascularization
- Exacerbation of <u>rheumatoid arthritis</u>

#### Reason:

To edit to correct text.

#### 12.9.2. Amendment 2 — Summary of Changes and Rationale

This is applicable to all study sites.

#### List of Protocol Changes with Rationale for Each

#### 1. PROTOCOL SYNOPSIS FOR STUDY PHI201754

#### **Analysis**

#### **Original Text:**

As a preliminary assessment, it will be confirmed if the mean Hgb in daprodustat group would lie fully within target range (10.0-12.0 g/dL) at first.

#### **Revised Text:**

As a preliminary assessment, it will be confirmed if the <u>lower and upper limit of 95% CI for</u> mean Hgb during the primary efficacy evaluation period in daprodustat group would lie fully within target range (10.0-12.0 g/dL) at first.

#### Reason:

To adjust description.

#### 1 PROTOCOL SYNOPSIS FOR STUDY PHI201754

#### Analysis

#### **Original Text:**

None

#### **Revised Text:**

Following sensitivity analyses will be conducted to assess robustness of study result.

- If there are Hgb considered to be impacted by blood transfusion or marketed rhEPO/ESAs, sensitivity analysis excluding the Hgb values from the analyses of primary endpoint will be conducted.
- Analysis of covariance (ANCOVA) will be conducted as sensitivity analysis to MMRM. This model includes treatment group and baseline Hgb. The analysis population will be mITT population and the similar analysis will be repeated in the PP population.
- A tipping point analysis based on multiple imputation will be conducted as sensitivity analysis to
  missing data assumption. This analysis explores a point where non-inferiority is not confirmed
  (tipping point) by changing assumption to missing data and repeating imputation. The analysis
  population will be ITT population and the similar analysis will be repeated in the mITT and PP
  population.

#### Reason:

To add sensitivity analyses for primary efficacy analyses and to adjust description.

#### **5.3.** Screening Failures

#### **Original Text:**

Screen failures are defined as subjects who consent to participate in the clinical trial <u>and are screened</u>, but are not subsequently officially enrolled in the study.

#### **Revised Text:**

Screen failures are defined as subjects who consent to participate in the clinical trial, but are not subsequently officially enrolled in the study.

#### Reason:

To change the definition of screening failures.

#### 5.4. Permanent discontinuation of study treatment and study withdrawal

#### **Original Text:**

• Need for chronic (more than 14 days) use of prohibited medication

#### **Revised Text:**

• Need for chronic (more than 14 days) use of prohibited medication (strong inhibitors/ inducers of CYP2C8 meet this criteria)

#### Reason:

To clarify discontinuation criteria (prohibited medication).

#### **6.9.** Treatment of Study Treatment Overdose

#### **Original Text:**

None

#### **Revised Text:**

For the purposes of this study, an overdose of daprodustat is defined as any dose greater than the highest daily dose included in the protocol.

#### Reason:

To clarify the definition of overdose of daprodustat.

#### 7.4.2. Adverse Events of Special Interest

#### **Original Text:**

 Death, myocardial infarction, stroke, <u>congestive</u> heart failure, <u>venous thromboembolism</u>, thrombosis of vascular access

#### **Revised Text:**

 Death, myocardial infarction, stroke, heart failure, <u>thromboembolic events</u>, thrombosis of vascular access

#### Reason:

To update AESI.

#### 9.1. Hypotheses

#### **Original Text:**

As a preliminary assessment, it will be confirmed whether the mean Hgb during the primary efficacy evaluation period in daprodustat group would be in target range (10.0-12.0 g/dL) at first.

#### **Revised Text:**

As a preliminary assessment, it will be confirmed whether the <u>lower and upper limit of 95% CI for</u> mean Hgb during the primary efficacy evaluation period in daprodustat group would be within target range (10.0-12.0 g/dL) at first.

#### Reason:

To adjust description.

#### 9.3.3. Adjustment for Multiplicity

#### **Original Text:**

Since the process will follow step-down manner, a multiplicity adjustment <u>for significance level of 5%</u> will not be needed according to a closed test procedure.

Other secondary endpoints, which will be evaluated on a complementary or exploratory basis, will be compared at a significance level of 5% without multiplicity adjustment.

#### **Revised Text:**

Since the process will follow step-down manner, a multiplicity adjustment will not be needed according to a closed test procedure, similarly two-sided significance level of 5% will be used. Other secondary endpoints, which will be evaluated on a complementary or exploratory basis, will be compared at a two-sided significance level of 5% without multiplicity adjustment.

#### Reason:

To adjust description.

#### 9.4.1. Primary Efficacy Analysis

#### **Original Text:**

None

#### **Revised Text:**

Following sensitivity analyses will be conducted to assess robustness of study result.

- If there are Hgb considered to be impacted by blood transfusion or marketed rhEPO/ESAs, sensitivity analysis excluding the Hgb values from the analyses of primary endpoint will be conducted.
- Analysis of covariance (ANCOVA) will be conducted as sensitivity analysis to MMRM. This model includes treatment group and baseline Hgb. The analysis population will be mITT population and the similar analysis will be repeated in the PP population.
- A tipping point analysis based on multiple imputation will be conducted as sensitivity analysis to missing data assumption. This analysis explores a point where non-inferiority is not confirmed (tipping point) by changing assumption to missing data and repeating imputation. The analysis population will be ITT population and the similar analysis will be repeated in the mITT and PP population.

#### Reason:

To add sensitivity analyses for primary efficacy analyses.

#### 12.1. Appendix 1: Abbreviations and Trademarks

**Trademark Information** 

Trademarks not owned by the GlaxoSmithKline group of companies

**Original Text:** 

None

#### **Revised Text:**

Nesp<sup>®</sup>

#### Reason:

To adjust description.

## 12.2. Appendix 2: Risk Assessment Potential Risk of Clinical Significance Original Text:

- - - -

Death, MI, stroke, <u>congestive</u> heart failure, <u>venous thromboembolism</u>, thrombosis of vascular access at Hgb levels which are within the normal range (i.e. not polycythemic conditions)

#### **Revised Text:**

Death, MI, stroke, heart failure, <u>thromboembolic events</u>, thrombosis of vascular access at Hgb levels which are within the normal range (i.e. not polycythemic conditions)

#### Reason:

To update summary of clinical significant potential risk.

PHI201754

# 12.2. Appendix 2: Risk Assessment Potential Risk of Clinical Significance Pulmonary artery hypertension (PAH) Summary of Data/Rationale for Risk Original Text:

Results from a clinical study of acute hypoxic challenge in healthy volunteers demonstrated that short-term therapy with daprodustat 5 mg or 10 mg has no clinically significant effect on echocardiographically estimated pulmonary artery systolic pressure (PASP) under either normoxic or hypoxic conditions.

#### **Revised Text:**

Results from a clinical study of acute hypoxic challenge in healthy volunteers demonstrated that short-term therapy with daprodustat 5 mg or 100 mg has no clinically significant effect on echocardiographically estimated pulmonary artery systolic pressure (PASP) under either normoxic or hypoxic conditions.

#### Reason:

To correct erroneous description.

#### 12.2. Appendix 2: Risk Assessment Potential Risk of Clinical Significance ESA risks (Control) Summary of Data/Rationale for Risk Original Text:

See risks outlined in table for daprodustat for Excessive erythropoiesis (polycythemia) leading to thrombosis and/or tissue ischemia; Risk of MI, stroke, <u>venous thromboembolism</u>, thrombosis of vascular access; and risk of cancer-related mortality and tumor progression.

#### **Revised Text:**

See risks outlined in table for daprodustat for Excessive erythropoiesis (polycythemia) leading to thrombosis and/or tissue ischemia; Risk of MI, stroke, <u>thromboembolic events</u>, thrombosis of vascular access; and risk of cancer-related mortality and tumor progression.

#### Reason:

To update summary of data/rationale for risk.